CLINICAL TRIAL: NCT02265952
Title: An Open-Label, Single-Arm, Proof-of-Concept Study to Evaluate the Safety and Efficacy of Single and Multiple Doses of REGN1500 in Patients With Homozygous Familial Hypercholesterolemia
Brief Title: Study of REGN1500 in Participants With Homozygous Familial Hypercholesterolemia (HoFH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R1500-CL-1331; 2016-000411-32 (EudraCT Number)
Record Dates: First submitted 2014-10-10; First posted 2014-10-16 (Estimated); Results first posted 2019-12-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Homozygous Familial Hypercholesterolemia
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia | interventions — evinacumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-label (Experimental): Open-label REGN1500
  Interventions: Drug: REGN1500 250 mg SC/15 mg/kg IV/450 mg SC

INTERVENTIONS:
Drug: REGN1500 250 mg SC/15 mg/kg IV/450 mg SC — Participants received single dose of REGN1500 subcutaneous (SC) injection of 250 milligrams (mg) at Week 0 (Day 1), followed by single dose of REGN1500 intravenous (IV) injection of 15 milligrams per kilogram (mg/kg) at Week 2 (Day 15) and then followed by 4 doses of REGN1500 SC injection of 450 mg once weekly starting from Week 12 (Day 85). Only the first 2 enrolled participants received 4 weekly REGN1500 450 mg SC doses at weeks 12, 13, 14, and 15 per the protocol. This dose regimen was removed under protocol amendment 4. Participants were followed for a period of 24 weeks (through Week 26 [Day 183]) after the last dose of study drug in the main study period.

SUMMARY:
This is an open-label, single-arm study to assess the reduction of low-density lipoprotein cholesterol (LDL-C) by REGN1500 in patients with homozygous familial hypercholesterolemia (HoFH).

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥18 years of age at the time of the screening visit
2. Diagnosis of homozygous familial hypercholesterolemia (HoFH)
3. Willing to consistently maintain usual diet for the duration of the study

Exclusion Criteria:

1. Background medical lipid modifying therapy that has not been stable for at least 4 weeks (6 weeks for fibrates) prior to the screening visit
2. Having undergone lipid apheresis within 4 weeks prior to the screening visit
3. Use of another investigational drug or therapy within 30 days or at least 5 half-lives (whichever is longer) prior to the screening visit
4. Previous participation in any clinical trial of REGN1500

Note: The information listed above is not intended to contain all considerations relevant to a patient's potential participation in this clinical trial therefore not all inclusion/ exclusion criteria are listed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-02-04 (Actual); Primary Completion 2016-11-21 (Actual); Study Completion 2018-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (5):
- United States (3):
  - Los Angeles, California
  - Philadelphia, Pennsylvania
  - Dallas, Texas
- Chicoutimi, Quebec, Canada
- Amsterdam, Netherlands

REFERENCES:
- [Background] Gaudet D, Gipe DA, Pordy R, Ahmad Z, Cuchel M, Shah PK, Chyu KY, Sasiela WJ, Chan KC, Brisson D, Khoury E, Banerjee P, Gusarova V, Gromada J, Stahl N, Yancopoulos GD, Hovingh GK. ANGPTL3 Inhibition in Homozygous Familial Hypercholesterolemia. N Engl J Med. 2017 Jul 20;377(3):296-297. doi: 10.1056/NEJMc1705994. No abstract available. PMID 28723334
- [Derived] Banerjee P, Chan KC, Tarabocchia M, Benito-Vicente A, Alves AC, Uribe KB, Bourbon M, Skiba PJ, Pordy R, Gipe DA, Gaudet D, Martin C. Functional Analysis of LDLR (Low-Density Lipoprotein Receptor) Variants in Patient Lymphocytes to Assess the Effect of Evinacumab in Homozygous Familial Hypercholesterolemia Patients With a Spectrum of LDLR Activity. Arterioscler Thromb Vasc Biol. 2019 Nov;39(11):2248-2260. doi: 10.1161/ATVBAHA.119.313051. Epub 2019 Oct 3. PMID 31578082

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at five sites in United States, Canada, and the Netherlands between 04 Feb 2015 and 23 Jul 2018. A total of 12 participants were screened in the study. Out of 12 participants, 9 participants received the study treatment.
Pre-assignment Details: This study consisted of 2 screening periods: 1st for main study and 2nd for open label extension (OLE) period. Participants on stable background medical lipid-modifying therapy for at least 4 weeks prior to screening, or who didn't undergo lipid apheresis within 4 weeks prior to screening visit, were directly entered into a 2-week screening period.
Groups:
- REGN1500 300 mg SC/20 mg/kg IV: Participants received REGN1500 SC injection of 300 mg at Week 26 (Day 183), 27(Day 190), 28 (Day 197) and 29 (Day 204) followed by IV injection of 20 mg/kg at Week 38 (Day 267) and every 12 weeks starting at Week 58 (Day 407) through Week 178 (Day 1247) in open-label extension period. Participants were to be followed for a period of 24 weeks (through Week 214 [Day 1499]) after the last dose of study drug in the OLE treatment period.
Period: Main Study Period
Arm/Group | REGN1500 250 mg SC/15 mg/kg IV/450 mg SC | REGN1500 300 mg SC/20 mg/kg IV
Started | 9 | 0
Completed | 9 | 0
Not Completed | 0 | 0
Period: Open Label Extension (OLE) Period
Arm/Group | REGN1500 250 mg SC/15 mg/kg IV/450 mg SC | REGN1500 300 mg SC/20 mg/kg IV
Started | 0 | 8
Completed | 0 | 0
Not Completed | 0 | 8
Not completed — Physician Decision | 0 | 7
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Arm/Group | REGN1500 250 mg SC/15 mg/kg IV/450 mg SC
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (9.06) [lower limit 9.06]
Age, Customized [Number; unit: Participants]
  < 45 years | 7
  ≥ 45 to < 65 years | 2
  ≥ 65 to < 75 years | 0
  < 75 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Ethnicity [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 6
  Not Reported | 0
Race [Count of Participants; unit: Participants]
  White | 7
  Black or African American | 0
  Asian | 0
  American Indian or Alaska Native | 0
  Native Hawaiian or Other Pacific Islander | 0
  Other | 0
  Not Reported | 2
Baseline Low-Density Lipoprotein Cholesterol (LDL-C) [Mean (Standard Deviation); unit: Milligram per Deciliter (mg/dL)] | 376.0 (240.85) [lower limit 240.85]
Baseline High-Density Lipoprotein Cholesterol (HDL-C) [Mean (Standard Deviation); unit: mg/dL] | 38.8 (14.24) [lower limit 14.24]
Baseline Non-High-Density Lipoprotein Cholesterol (Non-HDL-C) [Mean (Standard Deviation); unit: mg/dL] | 392.1 (246.41) [lower limit 246.41]
Baseline Apolipoprotein B (Apo B) [Mean (Standard Deviation); unit: mg/dL] | 226.1 (131.70) [lower limit 131.70]
Baseline Apolipoprotein CIII (Apo CIII) [Mean (Standard Deviation); unit: mg/dL] | 7.976 (3.3747) [lower limit 3.3747]
Baseline Triglyceride (TG) [Mean (Standard Deviation); unit: mg/dL] | 80.0 (41.20) [lower limit 41.20]
Baseline Lipoprotein(a) (Lp[a]) [Mean (Standard Deviation); unit: mg/dL] | 154.9 (109.25) [lower limit 109.25]
Baseline Total Cholesterol (Total -C) [Mean (Standard Deviation); unit: mg/dL] | 430.9 (235.60) [lower limit 235.60]
Baseline Apolipoprotein A-1 (Apo A-1) [Mean (Standard Deviation); unit: mg/dL] | 110.4 (23.74) [lower limit 23.74]

OUTCOME MEASURES:

1. Secondary Outcome: Absolute Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline (Week 0) to Week 4 in the Main Study Period
Description: Absolute change in low-density lipoprotein cholesterol (LDL-C) from baseline (week 0) up to week 4 was reported. The efficacy analysis set included all participants in the SAF who had baseline and at least 1 post-baseline measure of the lipid panel in the main study period.
Time Frame: Baseline (Week 0) up to Week 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | REGN1500 250 mg SC/15 mg/kg IV/450 mg SC
Number analyzed (Participants) | 9
mg/dL | -157.34 (89.590) [lower limit 89.590]

2. Primary Outcome: Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline (Week 0) to Week 4 in the Main Study Period
Description: Percent change was reported for low-density lipoprotein cholesterol (LDL-C) from baseline (week 0) up to week 4. LDL-C was measured using conventional units mg/dL. The efficacy analysis set included all participants in the safety analysis set (SAF) who had baseline and at least 1 post-baseline measure of the lipid panel in the main study period.
Time Frame: Baseline (Week 0) up to Week 4
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | REGN1500 250 mg SC/15 mg/kg IV/450 mg SC
Number analyzed (Participants) | 9
Percent Change | -49.17 (23.136) [lower limit 23.136]

3. Secondary Outcome: Absolute Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Week 2 to Week 4 in the Main Study Period
Description: Absolute change in low-density lipoprotein cholesterol (LDL-C) from week 2 to week 4 was reported. The efficacy analysis set included all participants in the SAF who had baseline and at least 1 post-baseline measure of the lipid panel in the main study period.
Time Frame: Week 2 to Week 4
Measure: Mean (Standard Deviation); unit: Milligram per Deciliter (mg/dL)
Arm/Group | REGN1500 250 mg SC/15 mg/kg IV/450 mg SC
Number analyzed (Participants) | 9
Milligram per Deciliter (mg/dL) | -63.63 (50.970) [lower limit 50.970]

4. Secondary Outcome: Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Week 2 to Week 4 in the Main Study Period
Description: Percent change was reported in low-density lipoprotein cholesterol (LDL-C) from week 2 to week 4. LDL-C was measured using conventional units mg/dL. The efficacy analysis set included all participants in the SAF who had baseline and at least 1 post-baseline measure of the lipid panel in the main study period.
Time Frame: Week 2 to Week 4
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | REGN1500 250 mg SC/15 mg/kg IV/450 mg SC
Number analyzed (Participants) | 9
Percent Change | -30.05 (18.503) [lower limit 18.503]

5. Secondary Outcome: Absolute Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline (Week 0) Over Time in the Main Study Period
Description: Absolute change was reported in low-density lipoprotein cholesterol (LDL-C) from baseline (week 0) up to week 26. The efficacy analysis set included all participants in the safety analysis set (SAF) who had baseline and at least 1 post-baseline measure of the lipid panel in the main study period.
Time Frame: Baseline (Week 0) up to Week 26
Population: "n" = Number of participants who were evaluable for this endpoint at a given time point.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | REGN1500 250 mg SC/15 mg/kg IV/450 mg SC
Number analyzed (Participants) | 9
mg/dL
  Change at Day 4 (n= 9) | -39.60 (41.677)
  Change at Week 1 (n= 9) | -67.59 (46.041)
  Change at Week 2 (n= 9) | -93.71 (86.504)
  Change at Week 3 (n= 9) | -129.97 (90.533)
  Change at Week 4 (n= 9) | -157.34 (89.590)
  Change at Week 5 (n= 8): number analyzed (Participants) | 8
  Change at Week 5 (n= 8) | -179.18 (101.260)
  Change at Week 6 (n= 9) | -183.41 (111.313)
  Change at Week 8 (n= 9) | -176.72 (118.441)
  Change at Week 10 (n= 9) | -151.19 (78.164)
  Change at Week 12 (n= 9) | -109.40 (74.108)
  Change at Week 13 (n= 2): number analyzed (Participants) | 2
  Change at Week 13 (n= 2) | -170.15 (105.288)
  Change at Week 14 (n= 9) | -104.16 (78.954)
  Change at Week 15 (n= 2): number analyzed (Participants) | 2
  Change at Week 15 (n= 2) | -186.15 (119.147)
  Change at Week 16 (n= 9) | -97.29 (179.016)
  Change at Week 17 (n= 2): number analyzed (Participants) | 2
  Change at Week 17 (n= 2) | -174.20 (103.803)
  Change at Week 18 (n= 7): number analyzed (Participants) | 7
  Change at Week 18 (n= 7) | -62.11 (167.004)
  Change at Week 20 (n= 2): number analyzed (Participants) | 2
  Change at Week 20 (n= 2) | -155.25 (79.832)
  Change at Week 22 (n= 7): number analyzed (Participants) | 7
  Change at Week 22 (n= 7) | -41.37 (169.432)
  Change at Week 23 (n= 2): number analyzed (Participants) | 2
  Change at Week 23 (n= 2) | -155.85 (78.984)
  Change at Week 25 (n= 2): number analyzed (Participants) | 2
  Change at Week 25 (n= 2) | -87.90 (23.900)
  Change at Week 26 (n= 6): number analyzed (Participants) | 6
  Change at Week 26 (n= 6) | -23.98 (152.794)

6. Secondary Outcome: Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline (Week 0) Over Time in the Main Study Period
Description: Percent change was reported in low-density lipoprotein cholesterol (LDL-C) from baseline (week 0) up to week 26. LDL-C was measured using conventional units mg/dL. The efficacy analysis set included all participants in the SAF who had baseline and at least 1 post-baseline measure of the lipid panel in the main study period.
Time Frame: Baseline (Week 0) up to Week 26
Population: "n" = Number of participants who were evaluable for this endpoint at a given time point.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | REGN1500 250 mg SC/15 mg/kg IV/450 mg SC
Number analyzed (Participants) | 9
Percent Change
  Percent change at Day 4 (n= 9) | -12.76 (11.086)
  Percent change at Week 1 (n= 9) | -24.00 (21.078)
  Percent change at Week 2 (n= 9) | -30.13 (24.402)
  Percent change at Week 3 (n= 9) | -41.38 (24.986)
  Percent change at Week 4 (n= 9) | -49.17 (23.136)
  Percent change at Week 5 (n= 8): number analyzed (Participants) | 8
  Percent change at Week 5 (n= 8) | -46.88 (14.507)
  Percent change at Week 6 (n= 9) | -52.13 (14.768)
  Percent change at Week 8 (n= 9) | -51.59 (17.910)
  Percent change at Week 10 (n= 9) | -45.61 (13.839)
  Percent change at Week 12 (n= 9) | -36.54 (19.281)
  Percent change at Week 13 (n= 2): number analyzed (Participants) | 2
  Percent change at Week 13 (n= 2) | -39.84 (10.753)
  Percent change at Week 14 (n= 9) | -33.02 (18.538)
  Percent change at Week 15 (n= 2): number analyzed (Participants) | 2
  Percent change at Week 15 (n= 2) | -43.38 (12.814)
  Percent change at Week 16 (n= 9) | -24.98 (25.441)
  Percent change at Week 17 (n= 2): number analyzed (Participants) | 2
  Percent change at Week 17 (n= 2) | -40.99 (9.950)
  Percent change at Week 18 (n= 7): number analyzed (Participants) | 7
  Percent change at Week 18 (n= 7) | -13.72 (28.424)
  Percent change at Week 20 (n= 2): number analyzed (Participants) | 2
  Percent change at Week 20 (n= 2) | -37.17 (5.503)
  Percent change at Week 22 (n= 7): number analyzed (Participants) | 7
  Percent change at Week 22 (n= 7) | -9.50 (38.456)
  Percent change at Week 23 (n= 2): number analyzed (Participants) | 2
  Percent change at Week 23 (n= 2) | -37.37 (5.217)
  Percent change at Week 25 (n= 2): number analyzed (Participants) | 2
  Percent change at Week 25 (n= 2) | -22.12 (2.537)
  Percent change at Week 26 (n= 6): number analyzed (Participants) | 6
  Percent change at Week 26 (n= 6) | -10.27 (25.806)

7. Secondary Outcome: Absolute Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline (Week 26) to Week 214 in the Open Label Extension (OLE) Period
Description: Absolute change in low-density lipoprotein cholesterol (LDL-C) from baseline (week 26) up to week 214 was reported. The efficacy analysis set included all participants in the SAF who had baseline and at least 1 post-baseline measure of the lipid panel in the main study period. (ET= Early Termination; EOS = End of Study)
Time Frame: Baseline (Week 26) up to Week 214
Population: "n" = Number of participants who were evaluable for this endpoint at a given time point.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | REGN1500 300 mg SC/20 mg/kg IV
Number analyzed (Participants) | 8
mg/dL
  Change at Week 26 (n= 8) | 261.34 (178.792)
  Change at Week 27 (n= 8) | -58.73 (56.992)
  Change at Week 28 (n= 8) | -88.16 (83.196)
  Change at Week 29 (n= 8) | -116.20 (102.219)
  Change at Week 30 (n= 7): number analyzed (Participants) | 7
  Change at Week 30 (n= 7) | -87.80 (108.905)
  Change at Week 31 (n= 8) | -144.99 (130.764)
  Change at Week 32 (n= 8) | -159.16 (128.072)
  Change at Week 34 (n= 8) | -128.38 (108.331)
  Change at Week 36 (n= 8) | -105.94 (89.990)
  Change at Week 38 (n= 8) | -79.98 (97.851)
  Change at Week 39 (n= 6): number analyzed (Participants) | 6
  Change at Week 39 (n= 6) | -138.28 (123.133)
  Change at Week 40 (n= 6): number analyzed (Participants) | 6
  Change at Week 40 (n= 6) | -127.13 (122.808)
  Change at Week 41 (n= 6): number analyzed (Participants) | 6
  Change at Week 41 (n= 6) | -163.28 (137.365)
  Change at Week 42 (n= 6): number analyzed (Participants) | 6
  Change at Week 42 (n= 6) | -142.65 (126.647)
  Change at Week 44 (n= 8) | -140.36 (109.275)
  Change at Week 46 (n= 8) | -123.25 (112.503)
  Change at Week 50 (n= 8) | -106.61 (99.458)
  Change at Week 54 (n= 8) | -13.38 (177.649)
  Change at Week 58 (n= 6): number analyzed (Participants) | 6
  Change at Week 58 (n= 6) | -48.27 (93.443)
  Change at Week 70 (n= 4): number analyzed (Participants) | 4
  Change at Week 70 (n= 4) | -117.93 (145.917)
  Change at Week 82 (n= 4): number analyzed (Participants) | 4
  Change at Week 82 (n= 4) | -63.88 (64.738)
  Change at Week 94 (n= 1): number analyzed (Participants) | 1
  Change at Week 94 (n= 1) | -369.90 (NA) — NA = Standard deviation cannot be calculated for n = 1.
  Change at Week 106 (n= 1): number analyzed (Participants) | 1
  Change at Week 106 (n= 1) | -290.00 (NA) — NA = Standard deviation cannot be calculated for n = 1.
  Change at ET (n= 8) | -9.78 (64.930)
  Change at EOS (n= 3): number analyzed (Participants) | 3
  Change at EOS (n= 3) | 95.63 (147.100)

8. Secondary Outcome: Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline (Week 26) to Week 214 in the Open Label Extension (OLE) Period
Description: Percent change was reported in low-density lipoprotein cholesterol (LDL-C) from baseline (week 26) to week 214 in the OLE period. LDL-C was measured using conventional units mg/dL. The efficacy analysis set included all participants in the SAF who had at least 1 post-baseline measure of the lipid panel in the main study period. (ET= Early Termination; EOS = End of Study)
Time Frame: Baseline (Week 26) up to Week 214
Population: "n" = Number of participants who were evaluable for this endpoint at a given time point.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | REGN1500 300 mg SC/20 mg/kg IV
Number analyzed (Participants) | 8
Percent Change
  Baseline (n= 8) | 261.34 (178.792)
  Percent change at Week 27 (n= 8) | -22.49 (16.520)
  Percent change at Week 28 (n= 8) | -36.74 (20.931)
  Percent change at Week 29 (n= 8) | -44.35 (20.817)
  Percent change at Week 30 (n= 7): number analyzed (Participants) | 7
  Percent change at Week 30 (n= 7) | -37.37 (31.297)
  Percent change at Week 31 (n= 8) | -50.74 (20.147)
  Percent change at Week 32 (n= 8) | -60.03 (18.502)
  Percent change at Week 34 (n= 8) | -53.03 (22.130)
  Percent change at Week 36 (n= 8) | -47.90 (21.623)
  Percent change at Week 38 (n= 8) | -37.05 (25.341)
  Percent change at Week 39 (n= 6): number analyzed (Participants) | 6
  Percent change at Week 39 (n= 6) | -59.83 (22.220)
  Percent change at Week 40 (n= 6): number analyzed (Participants) | 6
  Percent change at Week 40 (n= 6) | -53.90 (20.970)
  Percent change at Week 41 (n= 6): number analyzed (Participants) | 6
  Percent change at Week 41 (n= 6) | -66.28 (18.555)
  Percent change at Week 42 (n= 6): number analyzed (Participants) | 6
  Percent change at Week 42 (n= 6) | -59.59 (18.950)
  Percent change at Week 44 (n= 8) | -57.64 (18.599)
  Percent change at Week 46 (n= 8) | -48.74 (19.717)
  Percent change at Week 50 (n= 8) | -42.31 (23.194)
  Percent change at Week 54 (n= 8) | -13.60 (44.339)
  Percent change at Week 58 (n= 6): number analyzed (Participants) | 6
  Percent change at Week 58 (n= 6) | -12.86 (27.645)
  Percent change at Week 70 (n= 4): number analyzed (Participants) | 4
  Percent change at Week 70 (n= 4) | -38.61 (36.151)
  Percent change at Week 82 (n= 4): number analyzed (Participants) | 4
  Percent change at Week 82 (n= 4) | -24.68 (30.789)
  Percent change at Week 94 (n= 1): number analyzed (Participants) | 1
  Percent change at Week 94 (n= 1) | -81.67 (NA) — NA = Standard deviation cannot be calculated for n = 1.
  Percent change at Week 106 (n= 1): number analyzed (Participants) | 1
  Percent change at Week 106 (n= 1) | -64.03 (NA) — NA = Standard deviation cannot be calculated for n = 1.
  Percent change at ET (n= 8) | -17.65 (28.813)
  Percent change at EOS (n= 3): number analyzed (Participants) | 3
  Percent change at EOS (n= 3) | 19.59 (40.976)

9. Secondary Outcome: Absolute Change in Apolipoprotein (Apo B), Non-High-Density Lipoprotein Cholesterol (Non-HDL-C), Total Cholesterol (Total-C), and Lipoprotein(a) (Lp[a]) From Baseline (Week 0) up to Week 26 in the Main Study Period
Description: Absolute change was reported for Apo B, Non-HDL-C, Total-C, and Lp(a) from baseline (week 0) up to Week 26. The efficacy analysis set included all participants in the SAF who had baseline and at least 1 post-baseline measure of the lipid panel in the main study period.
Time Frame: Baseline (Week 0) up to Week 26
Population: "n" = Number of participants who were evaluable for this endpoint at a given time point.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | REGN1500 250 mg SC/15 mg/kg IV/450 mg SC
Number analyzed (Participants) | 9
mg/dL
  Apo B: Change at Week 2 (n = 9) | -53.0 (56.29)
  Apo B: Change at Week 3 (n = 9) | -81.0 (54.97)
  Apo B: Change at Week 4 (n = 9) | -96.3 (56.01)
  Apo B: Change at Week 5 (n = 8): number analyzed (Participants) | 8
  Apo B: Change at Week 5 (n = 8) | -104.6 (61.43)
  Apo B: Change at Week 6 (n = 9) | -100.7 (71.12)
  Apo B: Change at Week 8 (n = 9) | -96.8 (67.36)
  Apo B: Change at Week 12 (n = 9) | -60.0 (63.61)
  Apo B: Change at Week 14 (n = 9) | -61.7 (64.18)
  Apo B: Change at Week 16 (n = 9) | -62.6 (98.77)
  Apo B: Change at Week 18 (n = 7): number analyzed (Participants) | 7
  Apo B: Change at Week 18 (n = 7) | -28.6 (80.58)
  Apo B: Change at Week 20 (n = 2): number analyzed (Participants) | 2
  Apo B: Change at Week 20 (n = 2) | -114.0 (67.88)
  Apo B: Change at Week 22 (n = 7): number analyzed (Participants) | 7
  Apo B: Change at Week 22 (n = 7) | -22.7 (77.82)
  Apo B: Change at Week 23 (n = 2): number analyzed (Participants) | 2
  Apo B: Change at Week 23 (n = 2) | -119.0 (79.20)
  Apo B: Change at Week 26 (n = 6): number analyzed (Participants) | 6
  Apo B: Change at Week 26 (n = 6) | -4.7 (68.52)
  Non-HDL-C: Change at Day 4 (n = 9) | -44.61 (42.322)
  Non-HDL-C: Change at Week 1 (n = 9) | -72.16 (46.480)
  Non-HDL-C: Change at Week 2 (n = 9) | -97.12 (88.026)
  Non-HDL-C: Change at Week 3 (n = 9) | -138.09 (91.574)
  Non-HDL-C: Change at Week 4 (n = 9) | -165.64 (93.130)
  Non-HDL-C: Change at Week 5 (n = 8): number analyzed (Participants) | 8
  Non-HDL-C: Change at Week 5 (n = 8) | -187.46 (104.826)
  Non-HDL-C: Change at Week 6 (n = 9) | -191.20 (116.337)
  Non-HDL-C: Change at Week 8 (n = 9) | -182.98 (121.701)
  Non-HDL-C: Change at Week 10 (n = 9) | -156.98 (81.636)
  Non-HDL-C: Change at Week 12 (n = 9) | -116.20 (77.582)
  Non-HDL-C: Change at Week 13 (n = 2): number analyzed (Participants) | 2
  Non-HDL-C: Change at Week 13 (n = 2) | -180.25 (116.178)
  Non-HDL-C: Change at Week 14 (n = 9) | -108.58 (83.773)
  Non-HDL-C: Change at Week 15 (n = 2): number analyzed (Participants) | 2
  Non-HDL-C: Change at Week 15 (n = 2) | -196.85 (135.270)
  Non-HDL-C: Change at Week 16 (n = 9) | -99.58 (186.796)
  Non-HDL-C: Change at Week 17 (n = 2): number analyzed (Participants) | 2
  Non-HDL-C: Change at Week 17 (n = 2) | -185.40 (114.834)
  Non-HDL-C: Change at Week 18 (n = 7): number analyzed (Participants) | 7
  Non-HDL-C: Change at Week 18 (n = 7) | -60.41 (169.805)
  Non-HDL-C: Change at Week 20 (n = 2): number analyzed (Participants) | 2
  Non-HDL-C: Change at Week 20 (n = 2) | -161.90 (85.843)
  Non-HDL-C: Change at Week 22 (n = 7): number analyzed (Participants) | 7
  Non-HDL-C: Change at Week 22 (n = 7) | -41.16 (175.121)
  Non-HDL-C: Change at Week 23 (n = 2): number analyzed (Participants) | 2
  Non-HDL-C: Change at Week 23 (n = 2) | -163.25 (85.065)
  Non-HDL-C: Change at Week 25 (n = 2): number analyzed (Participants) | 2
  Non-HDL-C: Change at Week 25 (n = 2) | -92.20 (29.981)
  Non-HDL-C: Change at Week 26 (n = 6): number analyzed (Participants) | 6
  Non-HDL-C: Change at Week 26 (n = 6) | -25.47 (156.948)
  Total-C: Change at Day 4 (n = 9) | -50.36 (41.860)
  Total-C: Change at Week 1 (n = 9) | -81.99 (46.513)
  Total-C: Change at Week 2 (n = 9) | -109.03 (86.365)
  Total-C: Change at Week 3 (n = 9) | -154.10 (86.927)
  Total-C: Change at Week 4 (n = 9) | -180.79 (87.304)
  Total-C: Change at Week 5 (n = 8): number analyzed (Participants) | 8
  Total-C: Change at Week 5 (n = 8) | -199.11 (98.202)
  Total-C: Change at Week 6 (n = 9) | -207.63 (107.187)
  Total-C: Change at Week 8 (n = 9) | -195.18 (113.993)
  Total-C: Change at Week 10 (n = 9) | -167.87 (76.914)
  Total-C: Change at Week 12 (n = 9) | -122.94 (76.104)
  Total-C: Change at Week 13 (n = 2): number analyzed (Participants) | 2
  Total-C: Change at Week 13 (n = 2) | -188.45 (113.349)
  Total-C: Change at Week 14 (n = 9) | -114.68 (84.082)
  Total-C: Change at Week 15 (n = 2): number analyzed (Participants) | 2
  Total-C: Change at Week 15 (n = 2) | -205.60 (136.047)
  Total-C: Change at Week 16 (n = 9) | -105.24 (186.103)
  Total-C: Change at Week 17 (n = 2): number analyzed (Participants) | 2
  Total-C: Change at Week 17 (n = 2) | -195.00 (111.157)
  Total-C: Change at Week 18 (n = 7): number analyzed (Participants) | 7
  Total-C: Change at Week 18 (n = 7) | -63.27 (166.911)
  Total-C: Change at Week 20 (n = 2): number analyzed (Participants) | 2
  Total-C: Change at Week 20 (n = 2) | -170.45 (78.135)
  Total-C: Change at Week 22 (n = 7): number analyzed (Participants) | 7
  Total-C: Change at Week 22 (n = 7) | -41.30 (174.597)
  Total-C: Change at Week 23 (n = 2): number analyzed (Participants) | 2
  Total-C: Change at Week 23 (n = 2) | -167.55 (80.539)
  Total-C: Change at Week 25 (n = 2): number analyzed (Participants) | 2
  Total-C: Change at Week 25 (n = 2) | -90.15 (26.234)
  Total-C: Change at Week 26 (n = 6): number analyzed (Participants) | 6
  Total-C: Change at Week 26 (n = 6) | -30.77 (156.736)
  Lp(a): Change at Week 2 (n = 9) | -22.4 (30.18)
  Lp(a): Change at Week 3 (n = 9) | -20.8 (30.11)
  Lp(a): Change at Week 4 (n = 9) | -21.1 (28.29)
  Lp(a): Change at Week 5 (n = 8): number analyzed (Participants) | 8
  Lp(a): Change at Week 5 (n = 8) | -30.1 (24.91)
  Lp(a): Change at Week 6 (n = 9) | -25.0 (31.40)
  Lp(a): Change at Week 8 (n = 9) | -28.9 (23.81)
  Lp(a): Change at Week 12 (n = 9) | -20.9 (16.30)
  Lp(a): Change at Week 14 (n = 9) | -22.3 (21.01)
  Lp(a): Change at Week 16 (n = 9) | -26.9 (38.97)
  Lp(a): Change at Week 18 (n = 7): number analyzed (Participants) | 7
  Lp(a): Change at Week 18 (n = 7) | -29.9 (29.27)
  Lp(a): Change at Week 20 (n = 2): number analyzed (Participants) | 2
  Lp(a): Change at Week 20 (n = 2) | -19.0 (46.67)
  Lp(a): Change at Week 22 (n = 7): number analyzed (Participants) | 7
  Lp(a): Change at Week 22 (n = 7) | -24.3 (37.53)
  Lp(a): Change at Week 23 (n = 2): number analyzed (Participants) | 2
  Lp(a): Change at Week 23 (n = 2) | -12.5 (19.09)
  Lp(a): Change at Week 26 (n = 6): number analyzed (Participants) | 6
  Lp(a): Change at Week 26 (n = 6) | -16.3 (37.90)

10. Secondary Outcome: Percent Change in Apolipoprotein (Apo B), Non-High-Density Lipoprotein Cholesterol (Non-HDL-C), Total Cholesterol (Total-C), and Lipoprotein(a) (Lp[a]) From Baseline (Week 0) up to Week 26 in the Main Study Period
Description: Percent change was reported for Apo B, Non-HDL-C, Total-C, and Lp(a) from baseline (week 0) up to week 26. Apo B, Non-HDL-C, Total-C, and Lp(a) were measured using conventional units mg/dL. The efficacy analysis set included all participants in the SAF who had baseline and at least 1 post-baseline measure of the lipid panel in the main study period.
Time Frame: Baseline (Week 0) up to Week 26
Population: "n" = Number of participants who were evaluable for this endpoint at a given time point.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | REGN1500 250 mg SC/15 mg/kg IV/450 mg SC
Number analyzed (Participants) | 9
Percent Change
  Apo B: Percent change at Week 2 (n = 9) | -24.38 (20.959)
  Apo B: Percent change at Week 3 (n = 9) | -38.63 (22.114)
  Apo B: Percent change at Week 4 (n = 9) | -45.89 (18.222)
  Apo B: Percent change at Week 5 (n = 8): number analyzed (Participants) | 8
  Apo B: Percent change at Week 5 (n = 8) | -42.28 (13.247)
  Apo B: Percent change at Week 6 (n = 9) | -43.12 (14.716)
  Apo B: Percent change at Week 8 (n = 9) | -42.66 (14.475)
  Apo B: Percent change at Week 12 (n = 9) | -29.47 (21.736)
  Apo B: Percent change at Week 14 (n = 9) | -27.42 (18.418)
  Apo B: Percent change at Week 16 (n = 9) | -21.60 (24.970)
  Apo B: Percent change at Week 18 (n = 7): number analyzed (Participants) | 7
  Apo B: Percent change at Week 18 (n = 7) | -7.63 (24.347)
  Apo B: Percent change at Week 20 (n = 2): number analyzed (Participants) | 2
  Apo B: Percent change at Week 20 (n = 2) | -39.32 (6.481)
  Apo B: Percent change at Week 22 (n = 7): number analyzed (Participants) | 7
  Apo B: Percent change at Week 22 (n = 7) | -8.07 (30.444)
  Apo B: Percent change at Week 23 (n = 2): number analyzed (Participants) | 2
  Apo B: Percent change at Week 23 (n = 2) | -40.29 (10.089)
  Apo B: Percent change at Week 26 (n = 6): number analyzed (Participants) | 6
  Apo B: Percent change at Week 26 (n = 6) | -2.03 (25.320)
  Non-HDL-C: Percent change at Day 4 (n = 9) | -13.61 (10.721)
  Non-HDL-C: Percent change at Week 1 (n = 9) | -24.12 (20.083)
  Non-HDL-C: Percent change at Week 2 (n = 9) | -29.61 (23.406)
  Non-HDL-C: Percent change at Week 3 (n = 9) | -41.62 (23.969)
  Non-HDL-C: Percent change at Week 4 (n = 9) | -48.91 (22.257)
  Non-HDL-C: Percent change at Week 5 (n = 8): number analyzed (Participants) | 8
  Non-HDL-C: Percent change at Week 5 (n = 8) | -46.61 (14.172)
  Non-HDL-C: Percent change at Week 6 (n = 9) | -51.49 (14.344)
  Non-HDL-C: Percent change at Week 8 (n = 9) | -50.65 (17.231)
  Non-HDL-C: Percent change at Week 10 (n = 9) | -44.80 (13.148)
  Non-HDL-C: Percent change at Week 12 (n = 9) | -36.40 (18.711)
  Non-HDL-C: Percent change at Week 13 (n = 2): number analyzed (Participants) | 2
  Non-HDL-C: Percent change at Week 13 (n = 2) | -39.84 (11.313)
  Non-HDL-C: Percent change at Week 14 (n = 9) | -32.71 (18.214)
  Non-HDL-C: Percent change at Week 15 (n = 2): number analyzed (Participants) | 2
  Non-HDL-C: Percent change at Week 15 (n = 2) | -43.09 (14.482)
  Non-HDL-C: Percent change at Week 16 (n = 9) | -24.22 (25.899)
  Non-HDL-C: Percent change at Week 17 (n = 2): number analyzed (Participants) | 2
  Non-HDL-C: Percent change at Week 17 (n = 2) | -41.21 (10.455)
  Non-HDL-C: Percent change at Week 18 (n = 7): number analyzed (Participants) | 7
  Non-HDL-C: Percent change at Week 18 (n = 7) | -12.70 (27.798)
  Non-HDL-C: Percent change at Week 20 (n = 2): number analyzed (Participants) | 2
  Non-HDL-C: Percent change at Week 20 (n = 2) | -36.71 (5.471)
  Non-HDL-C: Percent change at Week 22 (n = 7): number analyzed (Participants) | 7
  Non-HDL-C: Percent change at Week 22 (n = 7) | -9.43 (37.102)
  Non-HDL-C: Percent change at Week 23 (n = 2): number analyzed (Participants) | 2
  Non-HDL-C: Percent change at Week 23 (n = 2) | -37.10 (5.138)
  Non-HDL-C: Percent change at Week 25 (n = 2): number analyzed (Participants) | 2
  Non-HDL-C: Percent change at Week 25 (n = 2) | -21.86 (1.676)
  Non-HDL-C: Percent change at Week 26 (n = 6): number analyzed (Participants) | 6
  Non-HDL-C: Percent change at Week 26 (n = 6) | -9.99 (25.292)
  Total-C: Percent change at Day 4 (n = 9) | -13.18 (8.932)
  Total-C: Percent change at Week 1 (n = 9) | -23.23 (16.602)
  Total-C: Percent change at Week 2 (n = 9) | -29.14 (20.307)
  Total-C: Percent change at Week 3 (n = 9) | -40.81 (21.011)
  Total-C: Percent change at Week 4 (n = 9) | -46.95 (19.083)
  Total-C: Percent change at Week 5 (n = 8): number analyzed (Participants) | 8
  Total-C: Percent change at Week 5 (n = 8) | -45.43 (12.909)
  Total-C: Percent change at Week 6 (n = 9) | -50.68 (13.327)
  Total-C: Percent change at Week 8 (n = 9) | -48.29 (15.556)
  Total-C: Percent change at Week 10 (n = 9) | -42.15 (10.858)
  Total-C: Percent change at Week 12 (n = 9) | -33.48 (16.136)
  Total-C: Percent change at Week 13 (n = 2): number analyzed (Participants) | 2
  Total-C: Percent change at Week 13 (n = 2) | -38.98 (10.525)
  Total-C: Percent change at Week 14 (n = 9) | -29.66 (15.759)
  Total-C: Percent change at Week 15 (n = 2): number analyzed (Participants) | 2
  Total-C: Percent change at Week 15 (n = 2) | -42.01 (14.356)
  Total-C: Percent change at Week 16 (n = 9) | -23.51 (25.208)
  Total-C: Percent change at Week 17 (n = 2): number analyzed (Participants) | 2
  Total-C: Percent change at Week 17 (n = 2) | -40.59 (9.468)
  Total-C: Percent change at Week 18 (n = 7): number analyzed (Participants) | 7
  Total-C: Percent change at Week 18 (n = 7) | -12.65 (26.105)
  Total-C: Percent change at Week 20 (n = 2): number analyzed (Participants) | 2
  Total-C: Percent change at Week 20 (n = 2) | -36.28 (3.862)
  Total-C: Percent change at Week 22 (n = 7): number analyzed (Participants) | 7
  Total-C: Percent change at Week 22 (n = 7) | -7.73 (33.729)
  Total-C: Percent change at Week 23 (n = 2): number analyzed (Participants) | 2
  Total-C: Percent change at Week 23 (n = 2) | -35.50 (4.662)
  Total-C: Percent change at Week 25 (n = 2): number analyzed (Participants) | 2
  Total-C: Percent change at Week 25 (n = 2) | -19.82 (1.459)
  Total-C: Percent change at Week 26 (n = 6): number analyzed (Participants) | 6
  Total-C: Percent change at Week 26 (n = 6) | -10.05 (22.903)
  Lp(a): Percent change at Week 2 (n = 9) | -11.64 (20.323)
  Lp(a): Percent change at Week 3 (n = 9) | -12.25 (19.350)
  Lp(a): Percent change at Week 4 (n = 9) | -10.85 (24.465)
  Lp(a): Percent change at Week 5 (n = 8): number analyzed (Participants) | 8
  Lp(a): Percent change at Week 5 (n = 8) | -23.79 (17.908)
  Lp(a): Percent change at Week 6 (n = 9) | -17.12 (23.680)
  Lp(a): Percent change at Week 8 (n = 9) | -17.24 (17.764)
  Lp(a): Percent change at Week 12 (n = 9) | -13.09 (12.614)
  Lp(a): Percent change at Week 14 (n = 9) | -13.54 (10.151)
  Lp(a): Percent change at Week 16 (n = 9) | -16.93 (24.795)
  Lp(a): Percent change at Week 18 (n = 7): number analyzed (Participants) | 7
  Lp(a): Percent change at Week 18 (n = 7) | -19.61 (21.686)
  Lp(a): Percent change at Week 20 (n = 2): number analyzed (Participants) | 2
  Lp(a): Percent change at Week 20 (n = 2) | -19.72 (32.894)
  Lp(a): Percent change at Week 22 (n = 7): number analyzed (Participants) | 7
  Lp(a): Percent change at Week 22 (n = 7) | -10.37 (29.230)
  Lp(a): Percent change at Week 23 (n = 2): number analyzed (Participants) | 2
  Lp(a): Percent change at Week 23 (n = 2) | -10.62 (15.373)
  Lp(a): Percent change at Week 26 (n = 6): number analyzed (Participants) | 6
  Lp(a): Percent change at Week 26 (n = 6) | 3.46 (39.400)

11. Secondary Outcome: Absolute Change in Apolipoprotein (Apo B), Non-High-Density Lipoprotein Cholesterol (Non-HDL-C), Total Cholesterol (Total-C), and Lipoprotein(a) (Lp[a]) From Baseline (Week 26) to Week 214 in the Open Label Extension (OLE) Period
Description: Absolute changein Apo B, Non-HDL-C, Total-C, and Lp(a) from baseline to week 214 in open label extension (OLE) period. The efficacy analysis set included all participants in the SAF who had baseline and at least one post-baseline measure of the lipid panel in the main study period. (ET = Early Termination; EOS = End of Study)
Time Frame: Baseline (Week 26) up to Week 214
Population: "n" = Number of participants who were evaluable for this endpoint at a given time point.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | REGN1500 300 mg SC/20 mg/kg IV
Number analyzed (Participants) | 8
mg/dL
  Apo B: Change at Week 30 (n= 7): number analyzed (Participants) | 7
  Apo B: Change at Week 30 (n= 7) | -48.1 (61.41)
  Apo B: Change at Week 34 (n= 8) | -65.9 (58.96)
  Apo B: Change at Week 38 (n= 8) | -40.9 (56.34)
  Apo B: Change at Week 42 (n= 6): number analyzed (Participants) | 6
  Apo B: Change at Week 42 (n= 6) | -79.5 (71.19)
  Apo B: Change at Week 44 (n= 8) | -78.6 (58.93)
  Apo B: Change at Week 50 (n= 8) | -57.8 (50.82)
  Apo B: Change at Week 70 (n= 4): number analyzed (Participants) | 4
  Apo B: Change at Week 70 (n= 4) | -60.3 (78.24)
  Apo B: Change at Week 82 (n= 4): number analyzed (Participants) | 4
  Apo B: Change at Week 82 (n= 4) | -38.0 (35.66)
  Apo B: Change at Week 94 (n= 1): number analyzed (Participants) | 1
  Apo B: Change at Week 94 (n= 1) | -212.0 (NA) — NA = Standard deviation cannot be calculated for n = 1.
  Apo B: Change at Week 106 (n= 1): number analyzed (Participants) | 1
  Apo B: Change at Week 106 (n= 1) | -173.0 (NA) — NA = Standard deviation cannot be calculated for n = 1.
  Apo B: Change at ET (n= 8) | -3.5 (42.88)
  Apo B: Change at EOS (n= 3): number analyzed (Participants) | 3
  Apo B: Change at EOS (n= 3) | 65.0 (100.53)
  Non- HDL-C: Change at Week 27 (n= 8) | -65.06 (61.756)
  Non- HDL-C: Change at Week 28 (n= 8) | -95.65 (87.499)
  Non- HDL-C: Change at Week 29 (n= 8) | -122.94 (106.296)
  Non- HDL-C: Change at Week 30 (n= 7): number analyzed (Participants) | 7
  Non- HDL-C: Change at Week 30 (n= 7) | -94.33 (113.286)
  Non- HDL-C: Change at Week 31 (n= 8) | -152.98 (135.977)
  Non- HDL-C: Change at Week 32 (n= 8) | -166.94 (133.990)
  Non- HDL-C: Change at Week 34 (n= 8) | -133.69 (112.247)
  Non- HDL-C: Change at Week 36 (n= 8) | -111.06 (93.635)
  Non- HDL-C: Change at Week 38 (n= 8) | -84.16 (101.210)
  Non- HDL-C: Change at Week 39 (n= 6): number analyzed (Participants) | 6
  Non- HDL-C: Change at Week 39 (n= 6) | -146.35 (128.368)
  Non- HDL-C: Change at Week 40 (n= 6): number analyzed (Participants) | 6
  Non- HDL-C: Change at Week 40 (n= 6) | -134.50 (128.198)
  Non- HDL-C: Change at Week 41 (n= 6): number analyzed (Participants) | 6
  Non- HDL-C: Change at Week 41 (n= 6) | -171.25 (143.692)
  Non- HDL-C:Change at Week 42 (n= 6): number analyzed (Participants) | 6
  Non- HDL-C:Change at Week 42 (n= 6) | -150.28 (132.214)
  Non- HDL-C: Change at Week 44 (n= 8) | -149.00 (114.152)
  Non- HDL-C: Change at Week 46 (n= 8) | -129.99 (116.770)
  Non- HDL-C: Change at Week 50 (n= 8) | -110.83 (104.353)
  Non- HDL-C: Change at Week 54 (n= 8) | -14.79 (178.797)
  Non- HDL-C: Change at Week 58 (n= 6): number analyzed (Participants) | 6
  Non- HDL-C: Change at Week 58 (n= 6) | -49.13 (97.212)
  Non- HDL-C: Change at Week 70 (n= 4): number analyzed (Participants) | 4
  Non- HDL-C: Change at Week 70 (n= 4) | -121.83 (152.887)
  Non- HDL-C: Change at Week 82 (n= 4): number analyzed (Participants) | 4
  Non- HDL-C: Change at Week 82 (n= 4) | -69.00 (66.715)
  Non- HDL-C: Change at Week 94 (n= 1): number analyzed (Participants) | 1
  Non- HDL-C: Change at Week 94 (n= 1) | -388.10 (NA) — NA = Standard deviation cannot be calculated for n = 1.
  Non- HDL-C: Change at Week 106 (n= 1): number analyzed (Participants) | 1
  Non- HDL-C: Change at Week 106 (n= 1) | -303.10 (NA) — NA = Standard deviation cannot be calculated for n = 1.
  Non- HDL-C: Change at ET (n= 8) | -12.45 (64.513)
  Non- HDL-C: Change at EOS (n= 3): number analyzed (Participants) | 3
  Non- HDL-C: Change at EOS (n= 3) | 102.07 (153.301)
  Total-C: Change at Week 27 (n= 8) | -73.80 (60.737)
  Total-C: Change at Week 28 (n= 8) | -107.78 (83.051)
  Total-C: Change at Week 29 (n= 8) | -134.33 (102.667)
  Total-C: Change at Week 30 (n= 7): number analyzed (Participants) | 7
  Total-C: Change at Week 30 (n= 7) | -107.61 (109.689)
  Total-C: Change at Week 31 (n= 8) | -166.85 (130.925)
  Total-C: Change at Week 32 (n= 8) | -181.09 (130.048)
  Total-C: Change at Week 34 (n= 8) | -148.90 (106.534)
  Total-C: Change at Week 36 (n= 8) | -125.14 (89.065)
  Total-C: Change at Week 38 (n= 8) | -93.00 (99.558)
  Total-C: Change at Week 39 (n= 6): number analyzed (Participants) | 6
  Total-C: Change at Week 39 (n= 6) | -160.38 (125.452)
  Total-C: Change at Week 40 (n= 6): number analyzed (Participants) | 6
  Total-C: Change at Week 40 (n= 6) | -150.42 (124.695)
  Total-C: Change at Week 41 (n= 6): number analyzed (Participants) | 6
  Total-C: Change at Week 41 (n= 6) | -188.42 (141.249)
  Total-C: Change at Week 42 (n= 6): number analyzed (Participants) | 6
  Total-C: Change at Week 42 (n= 6) | -166.80 (128.247)
  Total-C: Change at Week 44 (n= 8) | -164.68 (110.222)
  Total-C: Change at Week 46 (n= 8) | -144.69 (110.682)
  Total-C: Change at Week 50 (n= 8) | -123.04 (99.299)
  Total-C: Change at Week 54 (n= 8) | -23.80 (180.982)
  Total-C: Change at Week 58 (n= 6): number analyzed (Participants) | 6
  Total-C: Change at Week 58 (n= 6) | -54.45 (97.160)
  Total-C: Change at Week 70 (n= 4): number analyzed (Participants) | 4
  Total-C: Change at Week 70 (n= 4) | -132.55 (152.664)
  Total-C: Change at Week 82 (n= 4): number analyzed (Participants) | 4
  Total-C: Change at Week 82 (n= 4) | -75.43 (67.802)
  Total-C: Change at Week 94 (n= 1): number analyzed (Participants) | 1
  Total-C: Change at Week 94 (n= 1) | -392.30 (NA) — NA = Standard deviation cannot be calculated for n = 1.
  Total-C: Change at Week 106 (n= 1): number analyzed (Participants) | 1
  Total-C: Change at Week 106 (n= 1) | -303.10 (NA) — NA = Standard deviation cannot be calculated for n = 1.
  Total-C: Change at ET (n= 8) | -20.38 (68.809)
  Total-C: Change at EOS (n= 3): number analyzed (Participants) | 3
  Total-C: Change at EOS (n= 3) | 100.40 (144.828)
  Lp(a): Change at Week 30 (n= 7): number analyzed (Participants) | 7
  Lp(a): Change at Week 30 (n= 7) | -9.0 (27.59)
  Lp(a): Change at Week 34 (n= 8) | -10.8 (24.00)
  Lp(a): Change at Week 38 (n= 8) | -16.0 (19.70)
  Lp(a): Change at Week 42 (n= 6): number analyzed (Participants) | 6
  Lp(a): Change at Week 42 (n= 6) | -0.8 (41.36)
  Lp(a): Change at Week 44 (n= 8) | 1.5 (37.73)
  Lp(a): Change at Week 50 (n= 8) | 11.6 (48.23)
  Lp(a): Change at Week 70 (n= 4): number analyzed (Participants) | 4
  Lp(a): Change at Week 70 (n= 4) | 36.8 (77.92)
  Lp(a): Change at Week 82 (n= 4): number analyzed (Participants) | 4
  Lp(a): Change at Week 82 (n= 4) | -5.3 (27.04)
  Lp(a): Change at Week 94 (n= 1): number analyzed (Participants) | 1
  Lp(a): Change at Week 94 (n= 1) | -18.0 (NA) — NA = Standard deviation cannot be calculated for n = 1.
  Lp(a): Change at Week 106 (n= 1): number analyzed (Participants) | 1
  Lp(a): Change at Week 106 (n= 1) | 39.0 (NA) — NA = Standard deviation cannot be calculated for n = 1.
  Lp(a): Change at Week ET (n= 8) | 11.6 (26.72)
  Lp(a): Change at EOS (n= 3): number analyzed (Participants) | 3
  Lp(a): Change at EOS (n= 3) | 18.3 (18.01)

12. Secondary Outcome: Percent Change in Apolipoprotein (Apo B), Non-High-Density Lipoprotein Cholesterol (Non-HDL-C), Total Cholesterol (Total-C), and Lipoprotein(a) (Lp[a]) From Baseline (Week 26) to Week 214 in the Open Label Extension (OLE) Period
Description: Percent change was reported in Apo B, Non-HDL-C, Total-C, and Lp(a) from baseline (week 26) up to week 214 in OLE Period. Apo B, Non-HDL-C, Total-C, and Lp(a) were measured using conventional units mg/dL. The efficacy analysis set included all participants in the SAF who had baseline and at least one post-baseline measure of the lipid panel in the main study period. (ET= Early Termination; EOS = End of Study)
Time Frame: Baseline (Week 26) up to Week 214
Population: "n" = Number of participants who were evaluable for this endpoint at a given time point.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | REGN1500 300 mg SC/20 mg/kg IV
Number analyzed (Participants) | 8
Percent change
  Apo B: Percent change at Week 30 (n= 7): number analyzed (Participants) | 7
  Apo B: Percent change at Week 30 (n= 7) | -30.59 (25.991)
  Apo B: Percent change at Week 34 (n= 8) | -41.27 (19.573)
  Apo B: Percent change at Week 38 (n= 8) | -29.02 (25.029)
  Apo B: Percent change at Week 42 (n= 6): number analyzed (Participants) | 6
  Apo B: Percent change at Week 42 (n= 6) | -50.90 (17.497)
  Apo B: Percent change at Week 44 (n= 8) | -48.59 (16.201)
  Apo B: Percent change at Week 50 (n= 8) | -36.68 (19.620)
  Apo B: Percent change at Week 70 (n= 4): number analyzed (Participants) | 4
  Apo B: Percent change at Week 70 (n= 4) | -33.44 (26.773)
  Apo B: Percent change at Week 82 (n= 4): number analyzed (Participants) | 4
  Apo B: Percent change at Week 82 (n= 4) | -24.87 (17.148)
  Apo B: Percent change at Week 94 (n= 1): number analyzed (Participants) | 1
  Apo B: Percent change at Week 94 (n= 1) | -77.09 (NA) — NA = Standard deviation cannot be calculated for n = 1.
  Apo B: Percent change at Week 106 (n= 1): number analyzed (Participants) | 1
  Apo B: Percent change at Week 106 (n= 1) | -62.91 (NA) — NA = Standard deviation cannot be calculated for n = 1.
  Apo B: Percent change at ET (n= 8) | -11.94 (25.708)
  Apo B: Percent change at EOS (n= 3): number analyzed (Participants) | 3
  Apo B: Percent change at EOS (n= 3) | 22.60 (38.988)
  Non- HDL-C: Percent change at Week 27 (n= 8) | -23.62 (15.342)
  Non- HDL-C: Percent change at Week 28 (n= 8) | -37.22 (19.207)
  Non- HDL-C: Percent change at Week 29 (n= 8) | -44.30 (19.766)
  Non- HDL-C: Percent change at Week 30 (n= 7): number analyzed (Participants) | 7
  Non- HDL-C: Percent change at Week 30 (n= 7) | -37.90 (29.133)
  Non- HDL-C: Percent change at Week 31 (n= 8) | -50.59 (19.285)
  Non- HDL-C: Percent change at Week 32 (n= 8) | -59.09 (18.200)
  Non- HDL-C: Percent change at Week 34 (n= 8) | -51.55 (21.112)
  Non- HDL-C: Percent change at Week 36 (n= 8) | -46.62 (20.797)
  Non- HDL-C: Percent change at Week 38 (n= 8) | -36.10 (24.473)
  Non- HDL-C: Percent change at Week 39 (n= 6): number analyzed (Participants) | 6
  Non- HDL-C: Percent change at Week 39 (n= 6) | -59.25 (21.381)
  Non- HDL-C: Percent change at Week 40 (n= 6): number analyzed (Participants) | 6
  Non- HDL-C: Percent change at Week 40 (n= 6) | -53.24 (20.135)
  Non- HDL-C: Percent change at Week 41 (n= 6): number analyzed (Participants) | 6
  Non- HDL-C: Percent change at Week 41 (n= 6) | -65.07 (18.375)
  Non- HDL-C: Percent change at Week 42 (n= 6): number analyzed (Participants) | 6
  Non- HDL-C: Percent change at Week 42 (n= 6) | -58.92 (18.287)
  Non- HDL-C: Percent change at Week 44 (n= 8) | -57.03 (17.675)
  Non- HDL-C: Percent change at Week 46 (n= 8) | -48.27 (18.674)
  Non- HDL-C: Percent change at Week 50 (n= 8) | -41.16 (22.284)
  Non- HDL-C: Percent change at Week 54 (n= 8) | -12.93 (42.412)
  Non- HDL-C: Percent change at Week 58 (n= 6): number analyzed (Participants) | 6
  Non- HDL-C: Percent change at Week 58 (n= 6) | -12.28 (26.060)
  Non- HDL-C: Percent change at Week 70 (n= 4): number analyzed (Participants) | 4
  Non- HDL-C: Percent change at Week 70 (n= 4) | -37.68 (35.771)
  Non- HDL-C: Percent change at Week 82 (n= 4): number analyzed (Participants) | 4
  Non- HDL-C: Percent change at Week 82 (n= 4) | -26.16 (27.153)
  Non- HDL-C: Percent change at Week 94 (n= 1): number analyzed (Participants) | 1
  Non- HDL-C: Percent change at Week 94 (n= 1) | -81.52 (NA) — NA = Standard deviation cannot be calculated for n = 1.
  Non- HDL-C: Percent change at Week 106 (n= 1): number analyzed (Participants) | 1
  Non- HDL-C: Percent change at Week 106 (n= 1) | -63.66 (NA) — NA = Standard deviation cannot be calculated for n = 1.
  Non- HDL-C: Percent change at ET (n= 8) | -17.65 (27.339)
  Non- HDL-C: Percent change at EOS (n= 3): number analyzed (Participants) | 3
  Non- HDL-C: Percent change at EOS (n= 3) | 19.98 (40.313)
  Total-C: Percent change at Week 27 (n= 8) | -22.24 (11.566)
  Total-C: Percent change at Week 28 (n= 8) | -34.78 (14.984)
  Total-C: Percent change at Week 29 (n= 8) | -40.57 (14.335)
  Total-C: Percent change at Week 30 (n= 7): number analyzed (Participants) | 7
  Total-C: Percent change at Week 30 (n= 7) | -36.37 (23.550)
  Total-C: Percent change at Week 31 (n= 8) | -48.83 (16.944)
  Total-C: Percent change at Week 32 (n= 8) | -55.05 (16.624)
  Total-C: Percent change at Week 34 (n= 8) | -48.67 (18.123)
  Total-C: Percent change at Week 36 (n= 8) | -44.16 (19.175)
  Total-C: Percent change at Week 38 (n= 8) | -33.29 (22.145)
  Total-C: Percent change at Week 39 (n= 6): number analyzed (Participants) | 6
  Total-C: Percent change at Week 39 (n= 6) | -54.40 (19.803)
  Total-C: Percent change at Week 40 (n= 6): number analyzed (Participants) | 6
  Total-C: Percent change at Week 40 (n= 6) | -50.13 (18.316)
  Total-C: Percent change at Week 41 (n= 6): number analyzed (Participants) | 6
  Total-C: Percent change at Week 41 (n= 6) | -60.87 (17.966)
  Total-C: Percent change at Week 42 (n= 6): number analyzed (Participants) | 6
  Total-C: Percent change at Week 42 (n= 6) | -54.88 (15.886)
  Total-C: Percent change at Week 44 (n= 8) | -53.41 (16.231)
  Total-C: Percent change at Week 46 (n= 8) | -46.06 (16.855)
  Total-C: Percent change at Week 50 (n= 8) | -39.04 (19.318)
  Total-C: Percent change at Week 54 (n= 8) | -12.82 (38.323)
  Total-C: Percent change at Week 58 (n= 6): number analyzed (Participants) | 6
  Total-C: Percent change at Week 58 (n= 6) | -13.78 (21.976)
  Total-C: Percent change at Week 70 (n= 4): number analyzed (Participants) | 4
  Total-C: Percent change at Week 70 (n= 4) | -36.63 (32.371)
  Total-C: Percent change at Week 82 (n= 4): number analyzed (Participants) | 4
  Total-C: Percent change at Week 82 (n= 4) | -23.09 (19.171)
  Total-C: Percent change at Week 94 (n= 1): number analyzed (Participants) | 1
  Total-C: Percent change at Week 94 (n= 1) | -77.50 (NA) — NA = Standard deviation cannot be calculated for n = 1.
  Total-C: Percent change at Week 106 (n= 1): number analyzed (Participants) | 1
  Total-C: Percent change at Week 106 (n= 1) | -59.88 (NA) — NA = Standard deviation cannot be calculated for n = 1.
  Total-C: Percent change at ET (n= 8) | -16.76 (25.085)
  Total-C: Percent change at EOS (n= 3): number analyzed (Participants) | 3
  Total-C: Percent change at EOS (n= 3) | 18.20 (33.900)
  Lp(a): Percent change at Week 30 (n= 7): number analyzed (Participants) | 7
  Lp(a): Percent change at Week 30 (n= 7) | -3.57 (24.610)
  Lp(a): Percent change at Week 34 (n= 8) | -6.43 (21.281)
  Lp(a): Percent change at Week 38 (n= 8) | -9.50 (14.429)
  Lp(a): Percent change at Week 42 (n= 6): number analyzed (Participants) | 6
  Lp(a): Percent change at Week 42 (n= 6) | -4.76 (24.227)
  Lp(a): Percent change at Week 44 (n= 8) | -5.13 (25.377)
  Lp(a): Percent change at Week 50 (n= 8) | 1.02 (29.756)
  Lp(a): Percent change at Week 70 (n= 4): number analyzed (Participants) | 4
  Lp(a): Percent change at Week 70 (n= 4) | 15.80 (36.280)
  Lp(a): Percent change at Week 82 (n= 4): number analyzed (Participants) | 4
  Lp(a): Percent change at Week 82 (n= 4) | -3.77 (16.168)
  Lp(a): Percent change at Week 94 (n= 1): number analyzed (Participants) | 1
  Lp(a): Percent change at Week 94 (n= 1) | -11.92 (NA) — NA = Standard deviation cannot be calculated for n = 1.
  Lp(a): Percent change at Week 106 (n= 1): number analyzed (Participants) | 1
  Lp(a): Percent change at Week 106 (n= 1) | 25.83 (NA) — NA = Standard deviation cannot be calculated for n = 1.
  Lp(a): Percent change at ET (n= 8) | 9.96 (21.597)
  Lp(a): Percent change at EOS (n= 3): number analyzed (Participants) | 3
  Lp(a): Percent change at EOS (n= 3) | 40.51 (39.616)

13. Secondary Outcome: Percentage of Participants Who Achieved Reduction in Low-Density Lipoprotein Cholesterol (LDL-C) of ≥ 25% From Baseline (Week 0) in the Main Study Period
Description: Percentage of participants who achieved reduction in low-density lipoprotein cholesterol (LDL-C) of greater than or equal to (≥) 25 percent (%) from baseline in the main study period was reported. The efficacy analysis set included all participants in the SAF who had baseline and at least 1 post-baseline measure of the lipid panel in the main study period.
Time Frame: Baseline (Week 0) up to Week 26
Measure: Number; unit: Percentage of participants
Arm/Group | REGN1500 250 mg SC/15 mg/kg IV/450 mg SC
Number analyzed (Participants) | 9
Percentage of participants | 100

14. Secondary Outcome: Percentage of Participants Who Achieved Reduction in Low-Density Lipoprotein Cholesterol (LDL-C) of ≥ 25% From Baseline (Week 26) in the Open Label Extension (OLE) Period
Description: Percentage of participants who achieved a reduction in low-density lipoprotein cholesterol (LDL-C) of ≥ 25% from baseline (week 26) to week 214 was reported. The efficacy analysis set included all participants in the SAF who had baseline and at least 1 post-baseline measure of the lipid panel in the main study period.
Time Frame: Baseline (Week 26) to Week 214
Measure: Number; unit: Percentage of participants
Arm/Group | REGN1500 300 mg SC/20 mg/kg IV
Number analyzed (Participants) | 8
Percentage of participants | 100

15. Secondary Outcome: Percentage of Participants Who Achieved Reduction in Low-Density Lipoprotein Cholesterol (LDL-C) of ≥ 50% From Baseline (Week 0) in the Main Study Period
Description: Percentage of participants who achieved a reduction in low-density lipoprotein cholesterol (LDL-C) of ≥ 50% from baseline (week 0) to week 26 was reported. The efficacy analysis set included all participants in the SAF who had baseline and at least 1 post-baseline measure of the lipid panel in the main study period.
Time Frame: Baseline (Week 0) to Week 26
Measure: Number; unit: Percentage of participants
Arm/Group | REGN1500 250 mg SC/15 mg/kg IV/450 mg SC
Number analyzed (Participants) | 9
Percentage of participants | 77.8

16. Secondary Outcome: Percentage of Participants Who Achieved Reduction in Low-Density Lipoprotein Cholesterol (LDL-C) of ≥ 50% From Baseline (Week 26) in the Open Label Extension (OLE) Period
Description: Percentage of participants who achieved reduction in low-density lipoprotein cholesterol (LDL-C) of ≥ 50% from baseline (week 26) in the OLE period was reported. The efficacy analysis set included all participants in the SAF who had baseline and at least 1 post-baseline measure of the lipid panel in the main study period.
Time Frame: Baseline (Week 26) up to Week 214
Measure: Number; unit: Percentage
Arm/Group | REGN1500 300 mg SC/20 mg/kg IV
Number analyzed (Participants) | 8
Percentage | 87.5

17. Secondary Outcome: Absolute Change in High-Density Lipoprotein Cholesterol (HDL-C), Triglycerides (TG), and Apolipoprotein A-1 (Apo A-1) From Baseline (Week 0) Over Time in the Main Study Period
Description: Absolute change was reported in HDL-C, TG, and Apo A-1 from baseline (week 0) up to week 26. The efficacy analysis set included all participants in the SAF who had baseline and at least one post-baseline measure of the lipid panel in the main study period.
Time Frame: Baseline (Week 0) up to Week 26
Population: "n" = Number of participants who were evaluable for this endpoint at a given time point.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | REGN1500 250 mg SC/15 mg/kg IV/450 mg SC
Number analyzed (Participants) | 9
mg/dL
  HDL-C: Change at Day 4 (n = 9) | -5.81 (4.789)
  HDL-C: Change at Week 1 (n = 9) | -9.92 (6.578)
  HDL-C: Change at Week 2 (n = 9) | -11.99 (7.351)
  HDL-C: Change at Week 3 (n = 9) | -16.02 (10.737)
  HDL-C: Change at Week 4 (n = 9) | -15.07 (10.792)
  HDL-C: Change at Week 5 (n = 8): number analyzed (Participants) | 8
  HDL-C: Change at Week 5 (n = 8) | -11.66 (8.442)
  HDL-C: Change at Week 6 (n = 9) | -16.46 (11.868)
  HDL-C: Change at Week 8 (n = 9) | -12.06 (11.334)
  HDL-C: Change at Week 10 (n = 9) | -10.94 (8.215)
  HDL-C: Change at Week 12 (n = 9) | -6.82 (6.811)
  HDL-C: Change at Week 13 (n = 2): number analyzed (Participants) | 2
  HDL-C: Change at Week 13 (n = 2) | -8.10 (2.970)
  HDL-C: Change at Week 14 (n = 9) | -6.18 (4.205)
  HDL-C: Change at Week 15 (n = 2): number analyzed (Participants) | 2
  HDL-C: Change at Week 15 (n = 2) | -8.70 (0.566)
  HDL-C: Change at Week 16 (n = 9) | -5.54 (5.785)
  HDL-C: Change at Week 17 (n = 2): number analyzed (Participants) | 2
  HDL-C: Change at Week 17 (n = 2) | -9.40 (3.818)
  HDL-C: Change at Week 18 (n = 7): number analyzed (Participants) | 7
  HDL-C: Change at Week 18 (n = 7) | -2.93 (7.435)
  HDL-C: Change at Week 20 (n = 2): number analyzed (Participants) | 2
  HDL-C: Change at Week 20 (n = 2) | -8.70 (8.202)
  HDL-C: Change at Week 22 (n = 7): number analyzed (Participants) | 7
  HDL-C: Change at Week 22 (n = 7) | -0.30 (6.943)
  HDL-C: Change at Week 23 (n = 2): number analyzed (Participants) | 2
  HDL-C: Change at Week 23 (n = 2) | -4.00 (4.384)
  HDL-C: Change at Week 25 (n = 2): number analyzed (Participants) | 2
  HDL-C: Change at Week 25 (n = 2) | 2.50 (3.818)
  HDL-C: Change at Week 26 (n = 6): number analyzed (Participants) | 6
  HDL-C: Change at Week 26 (n = 6) | -5.30 (5.266)
  TG: Change at Day 4 (n = 9) | -25.17 (18.545)
  TG: Change at Week 1 (n = 9) | -21.41 (17.603)
  TG: Change at Week 2 (n = 9) | -15.83 (15.908)
  TG: Change at Week 3 (n = 9) | -39.73 (31.977)
  TG: Change at Week 4 (n = 9) | -40.81 (30.277)
  TG: Change at Week 5 (n = 8): number analyzed (Participants) | 8
  TG: Change at Week 5 (n = 8) | -42.04 (28.887)
  TG: Change at Week 6 (n = 9) | -38.73 (35.120)
  TG: Change at Week 8 (n = 9) | -30.37 (26.383)
  TG: Change at Week 10 (n = 9) | -28.79 (21.095)
  TG: Change at Week 12 (n = 9) | -33.23 (32.901)
  TG: Change at Week 13 (n = 2): number analyzed (Participants) | 2
  TG: Change at Week 13 (n = 2) | -49.15 (56.922)
  TG: Change at Week 14 (n = 9) | -22.11 (35.348)
  TG: Change at Week 15 (n = 2): number analyzed (Participants) | 2
  TG: Change at Week 15 (n = 2) | -52.20 (82.590)
  TG: Change at Week 16 (n = 9) | -11.20 (48.136)
  TG: Change at Week 17 (n = 2): number analyzed (Participants) | 2
  TG: Change at Week 17 (n = 2) | -55.35 (58.195)
  TG: Change at Week 18 (n = 7): number analyzed (Participants) | 7
  TG: Change at Week 18 (n = 7) | 9.77 (24.537)
  TG: Change at Week 20 (n = 2): number analyzed (Participants) | 2
  TG: Change at Week 20 (n = 2) | -33.65 (33.729)
  TG: Change at Week 22 (n = 7): number analyzed (Participants) | 7
  TG: Change at Week 22 (n = 7) | 1.90 (33.916)
  TG: Change at Week 23 (n = 2): number analyzed (Participants) | 2
  TG: Change at Week 23 (n = 2) | -36.30 (31.254)
  TG: Change at Week 25 (n = 2): number analyzed (Participants) | 2
  TG: Change at Week 25 (n = 2) | -23.45 (34.436)
  TG: Change at Week 26 (n = 6): number analyzed (Participants) | 6
  TG: Change at Week 26 (n = 6) | -5.87 (28.748)
  Apo A-1: Change at Week 2 (n = 9) | -28.6 (18.64)
  Apo A-1: Change at Week 3 (n = 9) | -43.3 (22.54)
  Apo A-1: Change at Week 4 (n = 9) | -43.4 (16.88)
  Apo A-1: Change at Week 5 (n = 8): number analyzed (Participants) | 8
  Apo A-1: Change at Week 5 (n = 8) | -35.8 (17.53)
  Apo A-1: Change at Week 6 (n = 9) | -40.7 (19.86)
  Apo A-1: Change at Week 8 (n = 9) | -33.6 (20.64)
  Apo A-1: Change at Week 12 (n = 9) | -17.2 (20.04)
  Apo A-1: Change at Week 14 (n = 9) | -17.7 (11.97)
  Apo A-1: Change at Week 16 (n = 9) | -11.3 (16.50)
  Apo A-1: Change at Week 18 (n = 7): number analyzed (Participants) | 7
  Apo A-1: Change at Week 18 (n = 7) | -4.9 (17.72)
  Apo A-1: Change at Week 20 (n = 2): number analyzed (Participants) | 2
  Apo A-1: Change at Week 20 (n = 2) | -24.0 (8.49)
  Apo A-1: Change at Week 22 (n = 7): number analyzed (Participants) | 7
  Apo A-1: Change at Week 22 (n = 7) | 1.9 (15.42)
  Apo A-1: Change at Week 23 (n = 2): number analyzed (Participants) | 2
  Apo A-1: Change at Week 23 (n = 2) | -23.0 (8.49)
  Apo A-1: Change at Week 26 (n = 6): number analyzed (Participants) | 6
  Apo A-1: Change at Week 26 (n = 6) | -10.8 (13.83)

18. Secondary Outcome: Percent Change in High-Density Lipoprotein Cholesterol (HDL-C), Triglycerides (TG), and Apolipoprotein A-1 (Apo A-1) From Baseline (Week 0) Over Time in the Main Study Period
Description: Percent change was reported in HDL-C, TG, and Apo A-1 from baseline (week 0) up to week 26. HDL-C, TG, and Apo A-1 were measured using conventional units mg/dL. The efficacy analysis set included all participants in the SAF who had baseline and at least 1 post-baseline measure of the lipid panel in the main study period.
Time Frame: Baseline (Week 0) up to Week 26
Population: "n" = Number of participants who were evaluable for this endpoint at a given time point.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | REGN1500 250 mg SC/15 mg/kg IV/450 mg SC
Number analyzed (Participants) | 9
Percent Change
  HDL-C: Percent Change at Day 4 (n = 9) | -14.37 (10.830)
  HDL-C: Percent Change at Week 1 (n = 9) | -23.34 (10.783)
  HDL-C: Percent Change at Week 2 (n = 9) | -28.75 (8.458)
  HDL-C: Percent Change at Week 3 (n = 9) | -36.96 (16.495)
  HDL-C: Percent Change at Week 4 (n = 9) | -35.24 (16.212)
  HDL-C: Percent Change at Week 5 (n = 8): number analyzed (Participants) | 8
  HDL-C: Percent Change at Week 5 (n = 8) | -29.74 (14.240)
  HDL-C: Percent Change at Week 6 (n = 9) | -37.88 (15.864)
  HDL-C: Percent Change at Week 8 (n = 9) | -25.42 (23.199)
  HDL-C: Percent Change at Week 10 (n = 9) | -24.57 (22.409)
  HDL-C: Percent Change at Week 12 (n = 9) | -13.59 (23.189)
  HDL-C: Percent Change at Week 13 (n = 2): number analyzed (Participants) | 2
  HDL-C: Percent Change at Week 13 (n = 2) | -24.48 (6.243)
  HDL-C: Percent Change at Week 14 (n = 9) | -16.81 (14.822)
  HDL-C: Percent Change at Week 15 (n = 2): number analyzed (Participants) | 2
  HDL-C: Percent Change at Week 15 (n = 2) | -26.97 (4.895)
  HDL-C: Percent Change at Week 16 (n = 9) | -12.03 (16.026)
  HDL-C: Percent Change at Week 17 (n = 2): number analyzed (Participants) | 2
  HDL-C: Percent Change at Week 17 (n = 2) | -28.34 (8.393)
  HDL-C: Percent Change at Week 18 (n = 7): number analyzed (Participants) | 7
  HDL-C: Percent Change at Week 18 (n = 7) | -1.05 (24.171)
  HDL-C: Percent Change at Week 20 (n = 2): number analyzed (Participants) | 2
  HDL-C: Percent Change at Week 20 (n = 2) | -25.39 (22.187)
  HDL-C: Percent Change at Week 22 (n = 7): number analyzed (Participants) | 7
  HDL-C: Percent Change at Week 22 (n = 7) | 3.78 (20.466)
  HDL-C: Percent Change at Week 23 (n = 2): number analyzed (Participants) | 2
  HDL-C: Percent Change at Week 23 (n = 2) | -11.56 (12.094)
  HDL-C: Percent Change at Week 25 (n = 2): number analyzed (Participants) | 2
  HDL-C: Percent Change at Week 25 (n = 2) | 8.41 (12.698)
  HDL-C: Percent Change at Week 26 (n = 6): number analyzed (Participants) | 6
  HDL-C: Percent Change at Week 26 (n = 6) | -12.00 (11.109)
  TG: Percent Change at Day 4 (n = 9) | -29.61 (18.562)
  TG: Percent Change at Week 1 (n = 9) | -23.41 (20.150)
  TG: Percent Change at Week 2 (n = 9) | -17.19 (18.735)
  TG: Percent Change at Week 3 (n = 9) | -44.38 (19.223)
  TG: Percent Change at Week 4 (n = 9) | -46.57 (17.014)
  TG: Percent Change at Week 5 (n = 8): number analyzed (Participants) | 8
  TG: Percent Change at Week 5 (n = 8) | -44.49 (16.583)
  TG: Percent Change at Week 6 (n = 9) | -40.03 (26.830)
  TG: Percent Change at Week 8 (n = 9) | -30.69 (24.800)
  TG: Percent Change at Week 10 (n = 9) | -31.40 (16.697)
  TG: Percent Change at Week 12 (n = 9) | -35.38 (25.014)
  TG: Percent Change at Week 13 (n = 2): number analyzed (Participants) | 2
  TG: Percent Change at Week 13 (n = 2) | -35.11 (26.733)
  TG: Percent Change at Week 14 (n = 9) | -23.51 (28.335)
  TG: Percent Change at Week 15 (n = 2): number analyzed (Participants) | 2
  TG: Percent Change at Week 15 (n = 2) | -27.77 (55.240)
  TG: Percent Change at Week 16 (n = 9) | -6.70 (40.326)
  TG: Percent Change at Week 17 (n = 2): number analyzed (Participants) | 2
  TG: Percent Change at Week 17 (n = 2) | -42.09 (22.941)
  TG: Percent Change at Week 18 (n = 7): number analyzed (Participants) | 7
  TG: Percent Change at Week 18 (n = 7) | 23.13 (55.349)
  TG: Percent Change at Week 20 (n = 2): number analyzed (Participants) | 2
  TG: Percent Change at Week 20 (n = 2) | -26.30 (11.945)
  TG: Percent Change at Week 22 (n = 7): number analyzed (Participants) | 7
  TG: Percent Change at Week 22 (n = 7) | 8.86 (43.819)
  TG: Percent Change at Week 23 (n = 2): number analyzed (Participants) | 2
  TG: Percent Change at Week 23 (n = 2) | -30.58 (6.662)
  TG: Percent Change at Week 25 (n = 2): number analyzed (Participants) | 2
  TG: Percent Change at Week 25 (n = 2) | -13.62 (21.582)
  TG: Percent Change at Week 26 (n = 6): number analyzed (Participants) | 6
  TG: Percent Change at Week 26 (n = 6) | -1.60 (33.318)
  Apo A-1: Percent Change at Week 2 (n = 9) | -24.37 (12.794)
  Apo A-1: Percent Change at Week 3 (n = 9) | -36.47 (16.930)
  Apo A-1: Percent Change at Week 4 (n = 9) | -38.54 (8.906)
  Apo A-1: Percent Change at Week 5 (n = 8): number analyzed (Participants) | 8
  Apo A-1: Percent Change at Week 5 (n = 8) | -31.91 (11.491)
  Apo A-1: Percent Change at Week 6 (n = 9) | -34.72 (12.342)
  Apo A-1: Percent Change at Week 8 (n = 9) | -29.03 (14.765)
  Apo A-1: Percent Change at Week 12 (n = 9) | -11.85 (25.176)
  Apo A-1: Percent Change at Week 14 (n = 9) | -17.65 (13.824)
  Apo A-1: Percent Change at Week 16 (n = 9) | -9.86 (14.372)
  Apo A-1: Percent Change at Week 18 (n = 7): number analyzed (Participants) | 7
  Apo A-1: Percent Change at Week 18 (n = 7) | -1.16 (19.598)
  Apo A-1: Percent Change at Week 20 (n = 2): number analyzed (Participants) | 2
  Apo A-1: Percent Change at Week 20 (n = 2) | -22.15 (7.965)
  Apo A-1: Percent Change at Week 22 (n = 7): number analyzed (Participants) | 7
  Apo A-1: Percent Change at Week 22 (n = 7) | 4.21 (17.857)
  Apo A-1: Percent Change at Week 23 (n = 2): number analyzed (Participants) | 2
  Apo A-1: Percent Change at Week 23 (n = 2) | -21.22 (7.959)
  Apo A-1: Percent Change at Week 26 (n = 6): number analyzed (Participants) | 6
  Apo A-1: Percent Change at Week 26 (n = 6) | -9.68 (11.250)

19. Secondary Outcome: Percent Change in High-Density Lipoprotein Cholesterol (HDL-C), Triglycerides (TG), and Apolipoprotein A-1 (Apo A-1) From Baseline (Week 26) to Week 214 in the Open Label Extension (OLE) Period
Description: Percent change was reported in HDL-C, TG and Apo A-1 from baseline (week 26) up to week 214. HDL-C, TG and Apo A-1 were measured using conventional units mg/dL. The efficacy analysis set included all participants in the SAF who had baseline and at least one post-baseline measure of the lipid panel in the main study period. (ET= Early Termination; EOS = End of Study)
Time Frame: Baseline (Week 26) up to Week 214
Population: "n" = Number of participants who were evaluable for this endpoint at a given time point.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | REGN1500 300 mg SC/20 mg/kg IV
Number analyzed (Participants) | 8
Percent change
  HDL-C: Percent change at Week 27 (n= 8) | -21.47 (11.815)
  HDL-C: Percent change at Week 28 (n= 8) | -27.60 (11.485)
  HDL-C: Percent change at Week 29 (n= 8) | -26.51 (16.584)
  HDL-C: Percent change at Week 30 (n= 7): number analyzed (Participants) | 7
  HDL-C: Percent change at Week 30 (n= 7) | -27.57 (14.566)
  HDL-C: Percent change at Week 31 (n= 8) | -32.81 (18.939)
  HDL-C: Percent change at Week 32 (n= 8) | -32.72 (14.684)
  HDL-C: Percent change at Week 34 (n= 8) | -34.60 (15.971)
  HDL-C: Percent change at Week 36 (n= 8) | -31.14 (18.695)
  HDL-C: Percent change at Week 38 (n= 8) | -18.57 (15.411)
  HDL-C: Percent change at Week 39 (n= 6): number analyzed (Participants) | 6
  HDL-C: Percent change at Week 39 (n= 6) | -32.09 (16.062)
  HDL-C: Percent change at Week 40 (n= 6): number analyzed (Participants) | 6
  HDL-C: Percent change at Week 40 (n= 6) | -36.25 (9.327)
  HDL-C: Percent change at Week 41 (n= 6): number analyzed (Participants) | 6
  HDL-C: Percent change at Week 41 (n= 6) | -39.14 (13.804)
  HDL-C: Percent change at Week 42 (n= 6): number analyzed (Participants) | 6
  HDL-C: Percent change at Week 42 (n= 6) | -38.31 (10.670)
  HDL-C: Percent change at Week 44 (n= 8) | -37.01 (12.049)
  HDL-C: Percent change at Week 46 (n= 8) | -32.77 (13.829)
  HDL-C: Percent change at Week 50 (n= 8) | -25.17 (17.957)
  HDL-C: Percent change at Week 54 (n= 8) | -20.16 (18.657)
  HDL-C: Percent change at Week 58 (n= 6): number analyzed (Participants) | 6
  HDL-C: Percent change at Week 58 (n= 6) | -10.87 (14.194)
  HDL-C: Percent change at Week 70 (n= 4): number analyzed (Participants) | 4
  HDL-C: Percent change at Week 70 (n= 4) | -24.67 (15.473)
  HDL-C: Percent change at Week 82 (n= 4): number analyzed (Participants) | 4
  HDL-C: Percent change at Week 82 (n= 4) | -17.56 (10.574)
  HDL-C: Percent change at Week 94 (n= 1): number analyzed (Participants) | 1
  HDL-C: Percent change at Week 94 (n= 1) | -13.95 (NA) — NA = Standard deviation cannot be calculated for n = 1.
  HDL-C: Percent change at Week 106 (n= 1): number analyzed (Participants) | 1
  HDL-C: Percent change at Week 106 (n= 1) | 0.00 (NA) — NA = Standard deviation cannot be calculated for n = 1.
  HDL-C: Percent change at ET (n= 8) | -15.08 (21.569)
  HDL-C: Percent change at EOS (n= 3): number analyzed (Participants) | 3
  HDL-C: Percent change at EOS (n= 3) | -0.78 (27.385)
  Triglycerides: Percent change at Week 27 (n= 8) | -38.62 (26.036)
  Triglycerides: Percent change at Week 28 (n= 8) | -41.76 (27.247)
  Triglycerides: Percent change at Week 29 (n= 8) | -41.17 (18.721)
  Triglycerides: Percent change at Week 30 (n= 7): number analyzed (Participants) | 7
  Triglycerides: Percent change at Week 30 (n= 7) | -38.82 (23.649)
  Triglycerides: Percent change at Week 31 (n= 8) | -44.86 (28.212)
  Triglycerides: Percent change at Week 32 (n= 8) | -45.33 (23.671)
  Triglycerides: Percent change at Week 34 (n= 8) | -28.58 (23.643)
  Triglycerides: Percent change at Week 36 (n= 8) | -25.89 (36.606)
  Triglycerides: Percent change at Week 38 (n= 8) | -24.32 (25.386)
  Triglycerides: Percent change at Week 39 (n= 6): number analyzed (Participants) | 6
  Triglycerides: Percent change at Week 39 (n= 6) | -48.37 (26.457)
  Triglycerides: Percent change at Week 40 (n= 6): number analyzed (Participants) | 6
  Triglycerides: Percent change at Week 40 (n= 6) | -43.36 (26.527)
  Triglycerides: Percent change at Week 41 (n= 6): number analyzed (Participants) | 6
  Triglycerides: Percent change at Week 41 (n= 6) | -46.65 (25.386)
  Triglycerides: Percent change at Week 42 (n= 6): number analyzed (Participants) | 6
  Triglycerides: Percent change at Week 42 (n= 6) | -43.09 (29.631)
  Triglycerides: Percent change at Week 44 (n= 8) | -47.98 (35.076)
  Triglycerides: Percent change at Week 46 (n= 8) | -37.64 (26.234)
  Triglycerides: Percent change at Week 50 (n= 8) | -22.10 (27.247)
  Triglycerides: Percent change at Week 54 (n= 8) | -1.08 (30.518)
  Triglycerides: Percent change at Week 58 (n= 6): number analyzed (Participants) | 6
  Triglycerides: Percent change at Week 58 (n= 6) | 3.72 (25.130)
  Triglycerides: Percent change at Week 70 (n= 4): number analyzed (Participants) | 4
  Triglycerides: Percent change at Week 70 (n= 4) | -22.28 (31.761)
  Triglycerides: Percent change at Week 82 (n= 4): number analyzed (Participants) | 4
  Triglycerides: Percent change at Week 82 (n= 4) | -36.47 (9.998)
  Triglycerides: Percent change at Week 94 (n= 1): number analyzed (Participants) | 1
  Triglycerides: Percent change at Week 94 (n= 1) | -76.36 (NA) — NA = Standard deviation cannot be calculated for n = 1.
  Triglycerides: Percent change at Week 106 (n= 1): number analyzed (Participants) | 1
  Triglycerides: Percent change at Week 106 (n= 1) | -57.98 (NA) — NA = Standard deviation cannot be calculated for n = 1.
  Triglycerides: Percent change at ET (n= 8) | -14.52 (25.892)
  Triglycerides: Percent change at EOS (n= 3): number analyzed (Participants) | 3
  Triglycerides: Percent change at EOS (n= 3) | 30.98 (40.511)
  Apo A-1: Percent change at Week 30 (n= 7): number analyzed (Participants) | 7
  Apo A-1: Percent change at Week 30 (n= 7) | -27.20 (12.119)
  Apo A-1: Percent change at Week 34 (n= 8) | -29.05 (17.483)
  Apo A-1: Percent change at Week 38 (n= 8) | -11.79 (23.939)
  Apo A-1: Percent change at Week 42 (n= 6): number analyzed (Participants) | 6
  Apo A-1: Percent change at Week 42 (n= 6) | -35.47 (9.512)
  Apo A-1: Percent change at Week 44 (n= 8) | -34.28 (11.306)
  Apo A-1: Percent change at Week 50 (n= 8) | -21.01 (15.471)
  Apo A-1: Percent change at Week 70 (n= 4): number analyzed (Participants) | 4
  Apo A-1: Percent change at Week 70 (n= 4) | -25.28 (11.950)
  Apo A-1: Percent change at Week 82 (n= 4): number analyzed (Participants) | 4
  Apo A-1: Percent change at Week 82 (n= 4) | -18.98 (6.534)
  Apo A-1: Percent change at Week 94 (n= 1): number analyzed (Participants) | 1
  Apo A-1: Percent change at Week 94 (n= 1) | -22.45 (NA) — NA = Standard deviation cannot be calculated for n = 1.
  Apo A-1: Percent change at Week 106 (n= 1): number analyzed (Participants) | 1
  Apo A-1: Percent change at Week 106 (n= 1) | 3.06 (NA) — NA = Standard deviation cannot be calculated for n = 1.
  Apo A-1: Percent change at ET (n= 8) | -9.63 (25.308)
  Apo A-1: Percent change at EOS (n= 3): number analyzed (Participants) | 3
  Apo A-1: Percent change at EOS (n= 3) | 11.27 (25.093)

20. Secondary Outcome: Absolute Change in High-Density Lipoprotein Cholesterol (HDL-C), Triglycerides (TG), and Apolipoprotein A-1 (Apo A-1) From Baseline (Week 26) to Week 214 in the Open Label Extension (OLE) Period
Description: Absolute change was reported in HDL-C, TG and Apo A-1 from baseline (week 26) up to week 214. The efficacy analysis set included all participants in the SAF who had baseline and at least one post-baseline measure of the lipid panel in the main study period. (ET= Early Termination; EOS = End of Study)
Time Frame: Baseline (Week 26) up to Week 214
Population: "n" = Number of participants who were evaluable for this endpoint at a given time point.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | REGN1500 300 mg SC/20 mg/kg IV
Number analyzed (Participants) | 8
mg/dL
  HDL-C: Change at Week 27 (n= 8) | -8.78 (5.736)
  HDL-C: Change at Week 28 (n= 8) | -12.08 (7.244)
  HDL-C: Change at Week 29 (n= 8) | -11.44 (7.858)
  HDL-C: Change at Week 30 (n= 7): number analyzed (Participants) | 7
  HDL-C: Change at Week 30 (n= 7) | -13.29 (9.270)
  HDL-C: Change at Week 31 (n= 8) | -13.94 (8.655)
  HDL-C: Change at Week 32 (n= 8) | -14.11 (8.163)
  HDL-C: Change at Week 34 (n= 8) | -15.10 (9.167)
  HDL-C: Change at Week 36 (n= 8) | -14.14 (10.426)
  HDL-C: Change at Week 38 (n= 8) | -8.89 (7.513)
  HDL-C: Change at Week 39 (n= 6): number analyzed (Participants) | 6
  HDL-C: Change at Week 39 (n= 6) | -14.02 (8.023)
  HDL-C: Change at Week 40 (n= 6): number analyzed (Participants) | 6
  HDL-C: Change at Week 40 (n= 6) | -15.90 (7.171)
  HDL-C: Change at Week 41 (n= 6): number analyzed (Participants) | 6
  HDL-C: Change at Week 41 (n= 6) | -17.17 (8.262)
  HDL-C: Change at Week 42 (n= 6): number analyzed (Participants) | 6
  HDL-C: Change at Week 42 (n= 6) | -16.65 (7.148)
  HDL-C: Change at Week 44 (n= 8) | -15.83 (8.167)
  HDL-C: Change at Week 46 (n= 8) | -14.85 (10.173)
  HDL-C: Change at Week 50 (n= 8) | -12.25 (10.985)
  HDL-C: Change at Week 54 (n= 8) | -9.06 (9.107)
  HDL-C: Change at Week 58 (n= 6): number analyzed (Participants) | 6
  HDL-C: Change at Week 58 (n= 6) | -5.42 (6.058)
  HDL-C: Change at Week 70 (n= 4): number analyzed (Participants) | 4
  HDL-C: Change at Week 70 (n= 4) | -10.83 (10.448)
  HDL-C: Change at Week 82 (n= 4): number analyzed (Participants) | 4
  HDL-C: Change at Week 82 (n= 4) | -6.28 (2.655)
  HDL-C: Change at Week 94 (n= 1): number analyzed (Participants) | 1
  HDL-C: Change at Week 94 (n= 1) | -4.20 (NA) — NA = Standard deviation cannot be calculated for n = 1.
  HDL-C: Change at Week 106 (n= 1): number analyzed (Participants) | 1
  HDL-C: Change at Week 106 (n= 1) | 0.00 (NA) — NA = Standard deviation cannot be calculated for n = 1.
  HDL-C: Percent change at ET (n= 8) | -7.86 (8.258)
  HDL-C: Change at EOS (n= 3): number analyzed (Participants) | 3
  HDL-C: Change at EOS (n= 3) | -1.67 (10.698)
  Triglycerides: Change at Week 27 (n= 8) | -31.19 (28.590)
  Triglycerides: Change at Week 28 (n= 8) | -36.28 (30.630)
  Triglycerides: Change at Week 29 (n= 8) | -32.86 (25.188)
  Triglycerides: Change at Week 30 (n= 7): number analyzed (Participants) | 7
  Triglycerides: Change at Week 30 (n= 7) | -32.37 (30.475)
  Triglycerides: Change at Week 31 (n= 8) | -39.04 (30.169)
  Triglycerides: Change at Week 32 (n= 8) | -37.83 (30.808)
  Triglycerides: Change at Week 34 (n= 8) | -25.41 (26.559)
  Triglycerides: Change at Week 36 (n= 8) | -24.66 (28.139)
  Triglycerides: Change at Week 38 (n= 8) | -21.13 (25.190)
  Triglycerides: Change at Week 39 (n= 6): number analyzed (Participants) | 6
  Triglycerides: Change at Week 39 (n= 6) | -40.27 (32.803)
  Triglycerides: Change at Week 40 (n= 6): number analyzed (Participants) | 6
  Triglycerides: Change at Week 40 (n= 6) | -37.30 (33.559)
  Triglycerides: Change at Week 41 (n= 6): number analyzed (Participants) | 6
  Triglycerides: Change at Week 41 (n= 6) | -39.37 (33.251)
  Triglycerides: Change at Week 42 (n= 6): number analyzed (Participants) | 6
  Triglycerides: Change at Week 42 (n= 6) | -37.62 (33.724)
  Triglycerides: Change at Week 44 (n= 8) | -42.25 (32.682)
  Triglycerides: Change at Week 46 (n= 8) | -31.53 (28.209)
  Triglycerides: Change at Week 50 (n= 8) | -20.00 (27.720)
  Triglycerides: Change at Week 54 (n= 8) | -6.40 (26.869)
  Triglycerides: Change at Week 58 (n= 6): number analyzed (Participants) | 6
  Triglycerides: Change at Week 58 (n= 6) | -3.53 (21.753)
  Triglycerides: Change at Week 70 (n= 4): number analyzed (Participants) | 4
  Triglycerides: Change at Week 70 (n= 4) | -21.23 (35.614)
  Triglycerides: Change at Week 82 (n= 4): number analyzed (Participants) | 4
  Triglycerides: Change at Week 82 (n= 4) | -26.33 (21.457)
  Triglycerides: Change at Week 94 (n= 1): number analyzed (Participants) | 1
  Triglycerides: Change at Week 94 (n= 1) | -88.50 (NA) — NA = Standard deviation cannot be calculated for n = 1.
  Triglycerides: Change at Week 106 (n= 1): number analyzed (Participants) | 1
  Triglycerides: Change at Week 106 (n= 1) | -67.20 (NA) — NA = Standard deviation cannot be calculated for n = 1.
  Triglycerides: Change at ET (n= 8) | -11.71 (21.343)
  Triglycerides: Change at EOS (n= 3): number analyzed (Participants) | 3
  Triglycerides: Change at EOS (n= 3) | 30.67 (35.390)
  Apo A-1: Change at Week 30 (n= 7): number analyzed (Participants) | 7
  Apo A-1: Change at Week 30 (n= 7) | -34.4 (20.18)
  Apo A-1: Change at Week 34 (n= 8) | -35.1 (24.70)
  Apo A-1: Change at Week 38 (n= 8) | -18.0 (26.54)
  Apo A-1: Change at Week 42 (n= 6): number analyzed (Participants) | 6
  Apo A-1: Change at Week 42 (n= 6) | -43.7 (15.71)
  Apo A-1: Change at Week 44 (n= 8) | -39.4 (18.12)
  Apo A-1: Change at Week 50 (n= 8) | -26.9 (23.56)
  Apo A-1: Change at Week 70 (n= 4): number analyzed (Participants) | 4
  Apo A-1: Change at Week 70 (n= 4) | -30.3 (20.12)
  Apo A-1: Change at Week 82 (n= 4): number analyzed (Participants) | 4
  Apo A-1: Change at Week 82 (n= 4) | -21.0 (5.83)
  Apo A-1: Change at Week 94 (n= 1): number analyzed (Participants) | 1
  Apo A-1: Change at Week 94 (n= 1) | -22.0 (NA) — NA = Standard deviation cannot be calculated for n = 1.
  Apo A-1: Change at Week 106 (n= 1): number analyzed (Participants) | 1
  Apo A-1: Change at Week 106 (n= 1) | 3.0 (NA) — NA = Standard deviation cannot be calculated for n = 1.
  Apo A-1: Change at ET (n= 8) | -15.6 (24.34)
  Apo A-1: Change at EOS (n= 3): number analyzed (Participants) | 3
  Apo A-1: Change at EOS (n= 3) | 7.0 (24.98)

21. Secondary Outcome: Absolute Change in Apolipoprotein CIII (Apo CIII) From Baseline (Week 0) Over Time in the Main Study Period
Description: Absolute change was reported in Apo CIII from baseline (week 0) up to week 16. The efficacy analysis set included all participants in the SAF who had baseline and at least 1 post-baseline measure of the lipid panel in the main study period.
Time Frame: Baseline (Week 0) up to Week 16
Population: "n" = Number of participants who were evaluable for this endpoint at a given time point.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | REGN1500 250 mg SC/15 mg/kg IV/450 mg SC
Number analyzed (Participants) | 9
mg/dL
  Apo CIII: Change at Day 4 (n = 9) | -3.729 (1.6905)
  Apo CIII: Change at Week 1 (n = 9) | -4.296 (1.9829)
  Apo CIII: Change at Week 2 (n = 9) | -4.301 (2.2542)
  Apo CIII: Change at Week 5 (n = 8): number analyzed (Participants) | 8
  Apo CIII: Change at Week 5 (n = 8) | -6.000 (2.8541)
  Apo CIII: Change at Week 6 (n = 1): number analyzed (Participants) | 1
  Apo CIII: Change at Week 6 (n = 1) | -8.380 (NA) — NA = Standard deviation cannot be calculated for n = 1.
  Apo CIII: Change at Week 12 (n = 9) | -3.772 (2.8443)
  Apo CIII: Change at Week 14 (n = 9) | -3.866 (3.7327)
  Apo CIII: Change at Week 16 (n = 9) | -2.757 (4.4877)

22. Secondary Outcome: Percent Change in Apolipoprotein CIII (Apo CIII) From Baseline (Week 0) Over Time in the Main Study Period
Description: Percent change was reported in Apo CIII from baseline (week 0) up to week 16. Apo CIII was measured using conventional units mg/dL. The efficacy analysis set included all participants in the SAF who had baseline and at least one post-baseline measure of the lipid panel in the main study period.
Time Frame: Baseline (Week 0) to Week 16
Population: "n" = Number of participants who were evaluable for this endpoint at a given time point.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | REGN1500 250 mg SC/15 mg/kg IV/450 mg SC
Number analyzed (Participants) | 9
Percent Change
  Apo CIII: Percent Change at Day 4 (n = 9) | -46.59 (22.129)
  Apo CIII: Percent Change at Week 1 (n = 9) | -55.43 (18.541)
  Apo CIII: Percent Change at Week 2 (n = 9) | -56.57 (24.815)
  Apo CIII: Percent Change at Week 5 (n = 8): number analyzed (Participants) | 8
  Apo CIII: Percent Change at Week 5 (n = 8) | -75.44 (9.667)
  Apo CIII: Percent Change at Week 6 (n = 1): number analyzed (Participants) | 1
  Apo CIII: Percent Change at Week 6 (n = 1) | -91.48 (NA) — NA = Standard deviation cannot be calculated for n = 1.
  Apo CIII: Percent Change at Week 12 (n = 9) | -49.07 (25.517)
  Apo CIII: Percent Change at Week 14 (n = 9) | -40.67 (44.674)
  Apo CIII: Percent Change at Week 16 (n = 9) | -28.30 (54.676)

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) were collected from signature of the informed consent form up to the final visit (up to Day 183 in Main Study Period, and up to Day 1499 in Open-Label Extension Period,regardless of seriousness or relationship to investigational product.
Description: During the main study period, the safety analysis set (SAF) was defined as all enrolled participants who received at least 1 dose or part of a dose. For OLE, the SAF was defined as all enrolled participants who received at least 1 dose or part of a dose in the OLE period. The SAF in both study periods was based on the treatment received (as treated).
Groups:
- Main Study Period: REGN1500 250 mg SC/15 mg/kg IV/450 mg SC: Participants received single dose of REGN1500 subcutaneous (SC) injection of 250 milligrams (mg) at Week 0 (Day 1), followed by single dose of REGN1500 intravenous (IV) injection of 15 milligrams per kilogram (mg/kg) at Week 2 (Day 15) and then followed by 4 doses of REGN1500 SC injection of 450 mg once weekly starting from Week 12 (Day 85). Only the first 2 enrolled participants received 4 weekly REGN1500 450 mg SC doses at weeks 12, 13, 14, and 15 per the protocol. This dose regimen was removed under protocol amendment 4. Participants were followed for a period of 24 weeks (through Week 26 [Day 183]) after the last dose of study drug in the main study period.
- OLE Period: REGN1500 300 mg SC/20 mg/kg IV: Participants received REGN1500 a SC injection of 300 mg at Week 26 (Day 183), 27(Day 190), 28 (Day 197) and 29 (Day 204) followed by IV injection of 20 mg/kg at Week 38 (Day 267) and every 12 weeks starting at Week 58 (Day 407) through Week 178 (Day 1247) in open-label extension period. Participants were to be followed for a period of 24 weeks (through Week 214 [Day 1499]) after the last dose of study drug in the OLE treatment period.
Arm/Group | Main Study Period: REGN1500 250 mg SC/15 mg/kg IV/450 mg SC | OLE Period: REGN1500 300 mg SC/20 mg/kg IV
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/9 | 2/8
Other Adverse Events (participants affected / at risk) | 9/9 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Study Period: REGN1500 250 mg SC/15 mg/kg IV/450 mg SC (N=9) | OLE Period: REGN1500 300 mg SC/20 mg/kg IV (N=8)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Study Period: REGN1500 250 mg SC/15 mg/kg IV/450 mg SC (N=9) | OLE Period: REGN1500 300 mg SC/20 mg/kg IV (N=8)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Corneal opacity (Eye disorders) | 1 (1) | 0 (0)
Eye inflammation (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 4 (6)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (6) | 3 (5)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Injection site haematoma (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 2 (3) | 2 (2)
Injection site haemorrhage (General disorders) | 1 (2) | 0 (0)
Local swelling (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Food allergy (Immune system disorders) | 0 (0) | 1 (2)
Gastroenteritis (Infections and infestations) | 1 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (3) | 3 (4)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (2) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Crush injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (3) | 1 (2)
Crystal urine present (Investigations) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 4 (8)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper-Airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Generalised erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Flushing (Vascular disorders) | 1 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
At the time patients completed the main study, the open-label extension (OLE) study was not yet open to enrollment. Therefore, there was a lag of between 168 days to 586 days between the end of the main study and the start of the OLE study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.